Version: 5.0 Date: 16 Apr 2024

#### TITLE PAGE

### **Protocol Title:**

A Comparative Crossover Study on the Safety, Efficacy, and Patient Quality of Life Comparing PureWick<sup>TM</sup> System with an Established Comparator in the Home Setting for Incontinence Overnight

**Protocol Number: UCC-8007** 

**Version Number: 5.0** 

**Investigational Device:** PureWick<sup>TM</sup> System

**Study Type:** Post-Market

**Short Title:** PureWick<sup>TM</sup> At-Home Pilot Study

Sponsor Name: C. R. Bard, Inc., a subsidiary of Becton, Dickinson and Company

Legal Registered Address: C. R. Bard, Inc.

8195 Industrial Blvd. Covington, GA 30014

Legal European Representative: BDI Benelux

Hagelberg 2 2250 Olen Belgium

**Sponsor Contact:** SengDao VanMany

Senior Clinical Project Manager

75 N Fairway Drive Vernon Hills, IL 60061 sengdao.vanmany@bd.com

(847)362-9209 (w) (847)732-6839 (c)

**Regulatory Agency Identifier Number(s):** NCT05710718 (USA), IDRCB: 2023-A01727-38 (France)

## **Overall Rationale for the protocol version 5.0:**

Protocol revised to incorporate new Quality of Life questionnaires (PROMIS Sleep Disturbance and End of Study Participant Preference Survey).


**Revision History** 

| Revision History Version Number | Date | Type |
|---|---|---|
| 1.0 | 30 Jan 2023 | Original |
| 2.0 | 26 June 2023 | Protocol update to allow inclusion of up to two investigational sites in both France and the US; administrative updates to correct and clarify text. |
| 3.0 | 14 August 2023 | Changes incorporated based on recommendations from the National Competent authority ANSM during their review: • Added Estimated start and end date of the study • Added IDRCB number |
| 4.0 | 5 September 2023 | Changes incorporated based on recommendations from the leading French etic committee during their review: • Added an additional exclusion criteria: Participants under supervision of a legally authorized representative are excluded to participate in the UCC-8007 trial • Deletion of the possibility for the home nurses to conduct virtual visits instead of face-to-face visits at day 30 |
| 5.0 | 08 April 2024 | Changes incorporated based on recommendations to include the following questionnaires: |


| Validated English and |
|----------------------------------|
| French version of the |
| PROMIS Sleep |
| Disturbance |
| Questionnaire |
| <ul> <li>End of Study</li> </ul> |
| Participant Preference |
| Survey |
| · |


# SPONSOR PROTOCOL APPROVAL

| Signature below indicates approval of the protocol as written. | | | |
|---|---|---|---|
| Individual or<br>function | Name | Signature | Date |
| Medical Affairs<br>Team Representative | Danielle Redmond<br>Medical Science Liaison,<br>Urology and Critical Care | This documen<br>electronically<br>system | 0 |
| Study Statistician | Yanchang Zhang<br>Statistician, Global Clinical<br>Affairs | This documen<br>electronically<br>system | 0 |
| Regulatory Affairs | Jenny McKinnon<br>Manager, Regulatory Affairs<br>Urology and Critical Care | This documen<br>electronically<br>system | 0 |
| Clinical Affairs | SengDao VanMany<br>Senior Clinical Project<br>Manager<br>Urology and Critical Care | This documen<br>electronically<br>system | |
| Project Manager | Winfried Huesmann<br>Clinical Program Manager,<br>EMEA | This documen<br>electronically<br>system | 0 |


## PROTOCOL SIGNATURE PAGE

# **Investigator Responsibilities**

Agreed to by (Investigator):

- 1. Prior to participation in this study, the Investigator or Institution must sign the Clinical Study Agreement (CSA) and obtain written approval from the appropriate Institutional Review Board (IRB)/Ethics Committee (EC).
- 2. The Investigator must receive BD-sponsored training prior to site activation. The Investigator is responsible for ensuring that all Sub-Investigators and clinical staff are adequately trained prior to performing any data collection or study-related procedures.
- 3. The Principal Investigator shall ensure that the study is conducted in accordance with the study protocol, any modifications as requested by the IRB/EC, the signed CSA, the ethical principles of the Declaration of Helsinki, Good Clinical Practice (ICH E6) / ISO 14155), and applicable national/regional regulations and laws.
- 4. If applicable, ensure that written informed consent is obtained from each participant prior to the conduct of any study procedure, using the current IRB/EC approved Informed Consent Form.

I have read and understand the contents of this study protocol. I agree to follow and abide by the requirements set forth in this document. I agree to conduct the trial in accordance with the study protocol, the signed Clinical Study Agreement, the signed Investigator Agreement and Good Clinical Practice (GCP) as well as applicable FDA and ISO regulations (e.g., 21 CFR Parts 50, 54, 56 and 812; 21 CFR Part 812.28 (a) (1) (Good Clinical Practice); EU MDR (Council Regulation 2017/745 of 5 April 2017), MDCG guidelines, and applicable national and regional law and regulation. I agree to participate in BD-Sponsored training prior to performing any data collection or study-related procedures.

| Printed Name – Investigator |
|-----------------------------|
| Signature – Investigator |
| Site Number |
| Date |


| TITLE PAGE | 1 |
|--------------------------------------------------------|----|
| Abbreviations | 10 |
| 1.0 PROTOCOL SUMMARY | 12 |
| 1.1 Synopsis | 12 |
| 1.2 Schema | 19 |
| 1.3 Schedule of Activities | 20 |
| 2.0 INTRODUCTION | 23 |
| 2.1 Background | 23 |
| 2.3 Rationale | 24 |
| 2.4 Risk/Benefit Assessment | 24 |
| 2.5 Risk Assessment | 25 |
| 2.5.1 Benefit Assessment | 27 |
| 2.5.2 Overall Benefit: Risk Conclusion | 28 |
| 3.0 OBJECTIVES AND ENDPOINTS | 28 |
| 4.0 STUDY DESIGN | 29 |
| 4.1 Overall Design | 29 |
| 4.2 Scientific Rationale for Study Design | 30 |
| 4.3 Participant Input into Design. | 30 |
| 4.4 End of Study Definition | 30 |
| 5.0 STUDY POPULATION | 30 |
| 5.1 Inclusion Criteria | 31 |
| 5.2 Exclusion Criteria | 31 |
| 5.3 Lifestyle Considerations | 31 |
| 5.4 Screen Failures | 31 |
| 6.0 STUDY INTERVENTION(S) | 32 |
| 6.1 Investigational/Test Device | 32 |
| 6.2 Pre-placement Procedure | 32 |
| 6.3 Control Device/Standard of Care | 33 |
| 6.4 Pre-placement Procedure | 33 |
| 6.5 Ancillary Devices/Products | 34 |
| 6.6 Device Labeling | 34 |
| 6.7 Treatment Allocation and Measures to Minimize Bias | 35 |
| 6.8 Randomization | 35 |

9.1.2

9.1.3

9.1.4

| Protocol Number: UCC-8007 CONFIDE | NTIAL |
|---|---|
| 9.3 Relationship of Adverse Event to Device(s)/Procedure | 44 |
| 9.4 Reporting of Events | 46 |
| 9.5 Serious Health Threats | 47 |
| 9.6 Safety Committees | 48 |
| 9.7 Device Deficiencies | 48 |
| 10.0 STATISTICAL METHODS | 48 |
| 10.1 Overview of Study Design | 49 |
| 10.2 Sample Size Considerations | 49 |
| 10.3 Analysis Population | 49 |
| 10.4 General Considerations | 49 |
| 10.4.1 Handling of Missing Data | 49 |
| 10.4.2 Poolability of Data | 50 |
| 10.4.3 Multiplicity Control | 50 |
| 10.5 Primary Endpoint(s) | 50 |
| 10.6 Secondary Endpoint(s) | 50 |
| 10.6.1 Questionnaire Nocturia Quality of Life (N-QoL) | 50 |
| 10.6.2 Questionnaire PROMIS Sleep Disturbance | 51 |
| 10.6.3 Tolerability - Number of days of actual use | 51 |
| 10.6.4 Tolerability - Discontinuation rate due to device discomfort or inconvenience | 51 |
| 10.6.5 Comfort, Ease of Use and Confidence | 51 |
| 10.7 Tertiary/Exploratory Endpoint(s) | 51 |
| 10.8 Other Analyses | 51 |
| 10.9 Interim Analyses | 51 |
| 11.0 DATA COLLECTION AND RECORD MAINTENANCE | 51 |
| 11.1 Case Report Forms | 51 |
| 11.2 Source Documentation | 52 |
| 11.3 Data Management | 52 |
| 11.4 Record Retention | 52 |
| 12.0 QUALITY CONTROL AND ASSURANCE | 53 |
| 12.1 Control of Study Products | 53 |
| 12.2 Monitoring | 53 |
| 12.3 Audits and Inspections | 54 |
| 12.4 Protocol Deviations | 54 |
| 13.0 ADMINISTRATIVE REQUIREMENTS | 55 |


# **Abbreviations**

| ADE | Adverse Device Effect |
|--------|------------------------------------------------------------|
| AE | Adverse event |
| Bard | C. R. Bard, Inc. |
| BD | Becton Dickinson and Company |
| CFR | Code of Federal Regulations |
| CI | Confidence Interval |
| CMP | Clinical Monitoring Plan |
| CRF | Case Report/Record Form |
| CRO | Contract Research Organization |
| CV | Curriculum Vitae |
| DMP | Data Management Plan |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| FDA | Food and Drug Administration |
| FDAAA | FDA Amendments Act of 2007 |
| FEC | Female External Catheter |
| FUP | Female Urinary Pouch |
| FR | France |
| GCP | Good Clinical Practice |
| HIPAA | Health Insurance Portability and Accountability Act |
| IAD | Incontinence Associated Dermatitis |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| IRB/EC | Institutional or Independent Review Board/Ethics Committee |
| MDCG | Medical Device Coordination Group |
| MDR | Medical Device Regulation |
| NDA | Non-disclosure Agreement |
| NSR | Non-significant Risk |
| OAB | Overactive Bladder Syndrome |
| PI | Principal Investigator |
| PUCS | PureWick™ Urine Collection System |
| PW | PureWick™ Female External Catheter |
| N-QOL | Nocturia Quality of Life |
| QOL | Quality of Life |
| RCT | Randomized Control Trial |
| RMV | Routine Monitoring Visit |
| SADE | Serious Adverse Device Effect |
| SAE | Serious Adverse Event |
| SD | Standard Deviation |
| SIV | Site Initiation Visit |
| SFTP | Secure File Transfer Protocol |


| SoA | Schedule of Activities |
|-------|------------------------------------------|
| SOP | Standard Operating Procedure |
| TMF | Trial Master File |
| UADE | Unexpected Adverse Device Effect |
| UI | Urinary Incontinence |
| U.S. | United States |
| USADE | Unexpected Serious Adverse Device Effect |


# 1.0 PROTOCOL SUMMARY

# 1.1 Synopsis

| Protocol Title | A Comparative Crossover Study on the Safety, Efficacy, and Patient Quality of Life Comparing PureWick <sup>TM</sup> System with an Established Comparator Overnight in the Home Setting for Incontinence. | |
|---|---|---|
| Short Title | PureWick™ At-Home Pilot Study | |
| Rationale | The study will collect clinical and quality of life data from patients requiring urine output management overnight in the home setting, which will aid reimbursement in France and the United States (U.S.). This pilot will inform the sample size and the frequency of nursing visits for the future randomized control trial. | |
| Objectives and Endpoints | Objective(s) | Endpoint(s) |
| | Primary To compare efficacy and safety of PureWick <sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device | <ul> <li>Efficacy – Daily capture rate via bed pad weights and captured volume.</li> <li>Safety – Daily skin irritation score using the Draize Scale.</li> </ul> |


## Secondary

- To assess impact of PureWick<sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device on Nocturnal Incontinence related Quality of Life and Sleep
- Tolerability To assess the tolerance of PureWick<sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device over the expected duration of use
- To assess participant comfort and ease of use of PureWick™ System and Hollister® Female Urinary Pouch External Collection Device
- To assess participant preference between the PureWick™ System and Hollister® Female Urinary Pouch External Collection Device after study completion

## Secondary

- Nocturia Quality of Life (N-QOL) score collected at baseline and every 2 weeks during treatment
- PROMIS Sleep
   Disturbance score at
   baseline and every 7th
   day during treatment.
- Tolerability Number of days of actual use of both devices & Discontinuation rate attributed to the device's inconvenience or discomfort.
- Overall comfort and ease
   of use scores on a 5-point
   Likert scale (brief
   questionnaire) collected at
   the end of each treatment
   phase.
- Overall preference via end of study participant preference survey administered at study completion.

Design and Overview

In this prospective, open-label, crossover trial, approximately 30 women with Nocturnal Urinary

Protocol Number: UCC-8007


Incontinence requiring the use of diapers in bed will be 1:1 randomized to a treatment sequence using two devices (PureWick<sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device) and followed for approximately 10 weeks through 2 treatment phases. For purposes of this study, the PureWick <sup>TM</sup> System will be referenced to include the PureWick<sup>TM</sup> Female External Catheter used in conjunction with the PureWick<sup>TM</sup> Urine Collection System, including the tubing and the canister.

At the start of the study, participants will be consented and screened against inclusion/exclusion criteria. All subjects that have met all eligibility criteria will be assigned a treatment order. Participants will view the training video for the applicable product at the beginning of each treatment phase and have access to the Instructions for Use (IFU) to review. Participants will use the device assigned in treatment phase 1 overnight while sleeping for 4 weeks (28 days) before transitioning to the second assigned device in treatment phase 2.

The primary endpoints will evaluate safety (skin injury) and efficacy (capture rate). Safety will be evaluated using the Draize Scale and efficacy will be measured based on daily capture rate.

Nurses will visit daily to measure urine capture rate and to assess for skin irritation using the Draize Scale.

The secondary outcomes include participative evaluation of the therapy and self-reported changes using questionnaires and preference surveys: Nocturia Quality of Life (N-QOL) assessment evaluated at baseline (previous treatment) and every 14 days through completion of each treatment phase (4 weeks/ 28 day period), PROMIS Sleep Disturbance measured at baseline and every 7 days through completion of each treatment phase, surveys (comfort & ease of use) completed by users at the end of each 4-week period, and end of study participant preference survey collected at study completion.

Tolerability to be measured by number of days of actual use of both devices, and discontinuation rate attributed to the device's discomfort or inconvenience.

## Investigational Device

#### Test product(s):

 PureWick<sup>TM</sup> Female External Catheter (PWFX30) (U.S.) and (PWFX30E) (EU)


| Dute: 10 / hpr 202 / | |
|---|---|
| Protocol Title | A Comparative Crossover Study on the Safety, Efficacy, and Patient Quality of Life Comparing PureWick <sup>TM</sup> System with an Established Comparator Overnight in the Home Setting for Incontinence. |
| | • PureWick™ Urine Collection System (PW100, PW200) (U.S.) and (PW200E) (EU) |
| | For regulatory status, refer to Regulatory Status row below within this table. |
| | Reference/Comparator product(s): |
| | Marketed Device: Hollister® Female Urinary Pouch External Collection Device |
| | Ancillary Product(s): |
| | <ul> <li>PureWick™ replacement Kit (PWKIT03) (U.S.) and (PWKIT03E) (EU)</li> <li>Absorbent under-pads</li> <li>Medium/Large sealing plastic bags</li> <li>Medical Triangular Graduated Cylinders, 1000mL</li> <li>Weighing Scales</li> <li>Urine Collection Bags for Hollister FUP</li> <li>Urine Bag Holders</li> <li>Mesh underwear</li> <li>PPE (Gloves, Chux)</li> <li>Barrier Paste</li> <li>Wipes</li> <li>Micropore tape</li> <li>Hair trimmers/clippers</li> </ul> |


## **Participants**

Adult female participants currently using incontinence products at night (e.g., nocturnal enuresis, nocturia, mobility limitation) will be recruited for this study from the study site.

To best mimic potential users of the PureWick™ System, participants ≥18 years of age will be enrolled. It is desired that at least 90% of participants are ≥65 years of age. This study will enroll approximately 30 participants.

#### **Inclusion Criteria**

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

- 1. Adult Female Participants ≥18 years of age at the time of signing the informed consent.
- 2. Currently use diapers or equivalent at night for urine capture ("Change complet" (FR))
- 3. Willing to comply with all study procedures in this protocol.
- 4. Provision of signed and dated informed consent form.

# **Exclusion Criteria**

Participants are excluded from the study if any of the following criteria apply:

- 1. Has frequent episodes of bowel incontinence without a fecal management system in place; or
- 2. Has moderate to heavy menstruation and cannot use a tampon or menstrual cup; or
- 3. Has Urinary tract, vaginal or other chronic infections, active genital herpes; or
- 4. Has Urinary retention; or
- 5. Is agitated, combative, and/or uncooperative and may remove the external catheter or pouch; or
- 6. Has any wound, open lesion or irritation on the genitalia, perineum, or sacrum; or
- 7. Has any pre-existing neurological, psychiatric, or other condition that would confound quality of life assessment or would make it difficult to self-report on quality-of-life questionnaires in the opinion of the investigator; or
- 8. Is known to be pregnant at time of enrollment (for


| Date: 16 Apr 2024 | |
|---|---|
| Protocol Title | A Comparative Crossover Study on the Safety, Efficacy, and Patient Quality of Life Comparing PureWick <sup>TM</sup> System with an Established Comparator Overnight in the Home Setting for Incontinence. |
| | women of childbearing age); or 9. Any other condition that, in the opinion of the investigator, would preclude them from participating in the study. 10. Is under supervision of a legally authorized representative |
| Intervention(s)/Procedure(s) | The PI or designee/nurse defined by the Draize Skin Score will assess skin and determine readiness for each treatment phase. Participants assigned to both treatment arms will place and remove the FEC (female external catheter) or FUP (Female Urinary Pouch) after standardized teaching is completed on the first day of the treatment phase. Participants will use the device assigned in treatment phases 1 and 2 overnight while sleeping for 4 weeks (28 days). |
| | There will be a minimum washout period of 2 weeks (not to exceed 4 weeks) between treatment phases. |
| Investigational Sites | Approximately 2 sites in France and approximately 2 sites in the U.S. |
| Data Monitoring Committee | N/A |
| Regulatory Status | Post-Market, Non-significant risk PureWick <sup>TM</sup> System |
| | <ul> <li>Class I, non-sterile device, CE marked, currently marketed in Europe</li> <li>Class I, 510(k) exempt device currently marketed in the U.S.</li> </ul> |
| | This investigation will use the PureWick <sup>TM</sup> System for its intended purpose. |
| Trial Duration | Estimated start date: (First Patient In): 19 Sep 2023 Estimated end date (Final Clinical Study Report): October 2024 |


| Protocol Title | A Comparative Crossover Study on the Safety, Efficacy, and Patient Quality of Life Comparing PureWick <sup>TM</sup> System with an Established Comparator Overnight in the Home Setting for Incontinence. |
|---|---|
| Regulatory Agency Identifier<br>Number(s): | NCT05710718 (USA) IDRCB: 2023-A01727-38 (France) |

Protocol Number: UCC-8007

Version: 5.0

Date: 16 Apr 2024

# 1.2 Schema



<sup>\*</sup>NQOL, PROMIS, Preference & Ease of Use assessments and questionnaires. Will be administered for both treatment phase 1 and 2.

<sup>\*\*</sup>Study Preference interview will only occur after participants have completed the study.

Protocol Number: UCC-8007


# 1.3 Schedule of Activities

| | | Daily Study Home Visits | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening /<br>Enrollment | Ph 1<br>Baseline<br>Day 1 | Ph1<br>Day<br>2-14 | Ph1<br>Day 15 | Ph1<br>Day<br>16-28 | Ph1<br>Day 29 | Ph1<br>Day<br>30 | Washout<br>Day 29-42<br>(+14 days) | Ph2<br>Baseline<br>Day 1 | Ph2<br>Day<br>2-14 | Ph2<br>Day<br>15 | Ph2<br>Day<br>16-28 | Ph2<br>Day<br>29 | Ph2<br>Day<br>30 |
| Informed consent | X | | | | | | | | | | | | | |
| Inclusion and exclusion criteria | X | | | | | | | | | | | | | |
| Demography | X | | | | | | | | | | | | | |
| Medical history | X | | | | | | | | | | | | | |
| Katz ADL Index | X | | | | | | | | | | | | | |
| Participant ID Assignment and Randomization | X | | | | | | | | | | | | | |
| Introduction to<br>Home Nurses<br>(On site or Virtual) | X | | | | | | | | | | | | | |
| Visual Skin Assessment & Draize Scoring (Both site and Nurses) | | X | X | X | X | X | X | | X | X | X | X | X | X |
| Nurses Confirm<br>Study Supplies | | X | | | | | | | X | | | | | |
| Nurses Have<br>Participant<br>Complete N-QOL | | Х | | X* | | X* | | | Х | | X* | | X* | |

Protocol Number: UCC-8007

Version: 5.0

Date: 16 Apr 2024

| 10 / Apr 2024 | | Daily Study Home Visits | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening /<br>Enrollment | Ph 1<br>Baseline<br>Day 1 | Ph1<br>Day<br>2-14 | Ph1<br>Day 15 | Ph1<br>Day<br>16-28 | Ph1<br>Day 29 | Ph1<br>Day<br>30 | Washout<br>Day 29-42<br>(+14 days) | Ph2<br>Baseline<br>Day 1 | Ph2<br>Day<br>2-14 | Ph2<br>Day<br>15 | Ph2<br>Day<br>16-28 | Ph2<br>Day<br>29 | Ph2<br>Day<br>30 |
| Nurses Have<br>Participant<br>Complete<br>PROMIS Sleep | | X | X*<br>Day 8 | X*<br>Day 15 | X*<br>Day 22 | X*<br>Day 29 | | | X | X*<br>Day 8 | X*<br>Day 15 | X*<br>Day 22 | X*<br>Day 29 | |
| Nurses Conduct<br>Device Training<br>w/Participants | | X | | | | | | | X | | | | | |
| Nurses Pre-weigh<br>urine canister or<br>graduated cylinder | | X | | | | | | | X | | | | | |
| Nurses Pre-Weigh<br>Overnight Pads<br>and Mesh<br>underwear<br>(if applicable) | | X | X | X | X | | | | X | X | X | X | | |
| Participants wear investigational device | | X | X | X | X | | | | X | X | X | X | | |
| Nurses Measure<br>Urine Output | | | X | X | X | X | | | | X | X | X | X | |
| Nurses Post-Weigh<br>Overnight Pads<br>and Mesh<br>Underwear<br>(if applicable) | | | X | X | X | X | | | | X | X | X | X | |
| Participant<br>Completes<br>Preference Survey | | | | | | X* | | | | | | | X* | |

Protocol Number: UCC-8007

Version: 5.0

Date: 16 Apr 2024

| | | Daily Study Home Visits | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening /<br>Enrollment | Ph 1<br>Baseline<br>Day 1 | Ph1<br>Day<br>2-14 | Ph1<br>Day 15 | Ph1<br>Day<br>16-28 | Ph1<br>Day 29 | Ph1<br>Day<br>30 | Washout<br>Day 29-42<br>(+14 days) | Ph2<br>Baseline<br>Day 1 | Ph2<br>Day<br>2-14 | Ph2<br>Day<br>15 | Ph2<br>Day<br>16-28 | Ph2<br>Day<br>29 | Ph2<br>Day<br>30 |
| Participant<br>Completes End of<br>Study Preference<br>Survey | | | | | | | | | | | | | X* | |
| AE review (If applicable) | | <b>—</b> | | | | | | | | | | | | <b>&gt;</b> |
| SAE review<br>(If applicable) | | <del>-</del> | | | | | | | | | | | | <b>→</b> |
| Device<br>Deficiencies<br>(If applicable) | | <b>—</b> | | | | | | | | | | | | <b>→</b> |

<sup>\*</sup>To be completed per treatment schedule or upon treatment discontinuation, whichever comes first.


## 2.0 INTRODUCTION

The PureWick<sup>TM®</sup> Female External Catheter (PureWick<sup>TM</sup> FEC) is an external drainage device to address the need for an effective, non-invasive method of managing urine output in adult incontinent women. The device utilizes suction to drain urine away from the patient through tubing that is connected to a collection canister. PureWick<sup>TM</sup> FEC can use either wall suction (acute care setting) or a free-standing PureWick<sup>TM</sup> Urine Collection System (home setting/skilled nursing facility). In the U.S., PureWick<sup>TM</sup> FEC is a Class I, 510(k) exempt device. In Europe, the PureWick<sup>TM</sup> FEC is a Class I, CE marked, non-sterile device.

## 2.1 Background

Adult nocturnal enuresis, or nighttime urinary incontinence in the home setting has a significant impact on the individual, their family or caregiver, and the broader health system. Nocturnal enuresis in the adult population may be related to a multitude of causes, including but not limited to OAB (Overactive Bladder syndrome), dementia, mobility issues, and nocturia<sup>9</sup>. There is an apparent lack of research and focused attention on urinary incontinence management in people living at home.<sup>3</sup> With an aging population and the emerging acceptance of open discussion of urinary management needs, there is an urgent need for both research and products tailored to those living in their home, where most adults with nighttime incontinence live.<sup>3</sup>

Current literature supports that incontinence is under-reported. <sup>9,13</sup> One qualitative study looking at those with dementia and incontinence reported, "Most carers reported protecting the person's dignity by not seeking health professionals help often until the point of a crisis" and incontinent women were less likely to seek care for their incontinence compared with incontinent men. <sup>7</sup> Not only are patients and their caregivers embarrassed to discuss incontinence with their provider, but they're also embarrassed about the multiple challenges with available toileting supplies, <sup>4</sup> which has highlighted the need for urinary management solutions. In addition to being under-reported, older people frequently are not assessed and treated. <sup>13</sup>

Although prevalence reports range, urinary incontinence (UI) rates among women are consistently high, especially in the elderly. The burden of UI amongst elderly people in the United States (U.S.) is immense, with UI prevalence estimates for elderly community-dwelling women approximately 41% of Medicare beneficiaries <sup>11</sup> ranging up to 55%. <sup>10</sup> UI represents a similar public health burden in France, with 25% to 40% of women declaring suffering from UI and an increasing prevalence with age, with UI rates exceeding 45% among 75+ year-old women. <sup>28</sup>

Quality of Life (QOL) is impacted in women with UI,<sup>13</sup> including comorbidities and poorer health overall (despite education, poverty status, or smoking), including falls<sup>10</sup> and positive bacterial cultures in those with UI in nursing homes<sup>5</sup>, physical and mental health (independent of demographic factors and comorbidities).<sup>8</sup>, and Incontinence Associated Dermatitis (IAD).<sup>12</sup> These represent meaningful constraints in physical and social


activities, along with significant impacts on emotional well-being.<sup>6,8</sup> One potential solution discussed by an older eleven-site European research project is to empower elderly individuals with incontinence to stay in their own homes with a better quality of life is that they would require caregiver assistance during toileting regularly<sup>1</sup>, which adds additional expense. A recent Conjoint Analysis survey revealed that getting a good night's sleep and feeling rested were most important to individuals with nocturnal enuresis.<sup>24</sup>

Finally, incontinence correlated with a considerable economic burden from both a patient perspective and in the community. 14,16,17,18,19,20,21,22,23 In addition to direct costs, to be taken into consideration is the need to institutionalize loved ones because incontinence cannot be managed in the home setting. The ability to independently use the toilet and urinary incontinence appear to be independent predictors of the elderly and their families choosing admission to an institution. 15 Considering OAB alone, a retrospective study among Medicare beneficiaries indicated that the cost of care for female patients in nursing homes is higher than for female patients in nursing homes without OAB. 16 Estimates of the economic burden associated with OAB have been derived from community-dwelling populations. 9,12

Further research is needed to determine if there's an unmet need for current solutions to identified problems such as the need for additional caregivers or admission to institutions, Quality of Life solutions, or product alternatives that are safe and effective, and if there is potential to improve quality of life, or delay nursing home admissions with alternative home care solutions. A recently published patient and caregiver satisfaction survey with the PureWick<sup>TM</sup> System used in the home setting showed over 80% satisfaction, comfort, and ease of use using the product compared with their baseline incontinence solution despite over 70% reporting the PureWick<sup>TM</sup> System had a higher cost compared with their baseline direct costs.<sup>25</sup>

The PureWick<sup>TM</sup> Urine Collection System (PUCS) is to be used with PureWick<sup>TM</sup> External Catheters (FEC) which are intended for non-invasive urine output management and will be collectively referenced as the PureWick<sup>TM</sup> System throughout this study.

### 2.3 Rationale

The study will collect clinical and quality of life data from patients requiring urine output management overnight in the home setting, which will aid reimbursement in France and the United States (U.S.). This pilot will inform the sample size and the frequency of nursing visits for the future home-setting, randomized control trial.

#### 2.4 Risk/Benefit Assessment

Subjects participating in this study will be treated with approved, marketed devices and will use the investigational devices as intended. Therefore, subjects will be exposed to the same risks shared by all patients using these devices for urine output management in a real-world setting. More detailed information about the known and expected benefits and risks


and reasonably expected adverse events of the PureWick<sup>TM</sup> Female External Catheter, PureWick Urine Collection System and the Hollister® Female Urinary Pouch External Collection Device may be found in the Instructions for Use for each product.

# 2.5 Risk Assessment

| Potential Risk of Clinical Significance | Summary of<br>Data/Rationale for Risk | Mitigation Strategy |
|---|---|---|
| Study Intervention: PureWick <sup>TM</sup> System | | |
| Potential adverse events: Skin Injury Skin Irritation Allergic Reaction | PureWick <sup>TM</sup> FEC is an external device placed between the separated gluteus and labia; it is in direct contact with skin and mucous membranes | <ul> <li>To avoid potential skin injury, never push or pull the PureWick<sup>TM</sup> Female External Catheter against the skin during placement or removal.</li> <li>Assess local area before device application/after device removal and periodically throughout use.</li> <li>To monitor skin irritation, daily skin assessment will be performed using the Draize scale.</li> <li>To avoid allergic reactions, study is using Non-latex PureWick<sup>TM</sup> FEC</li> </ul> |
| Potential adverse events: | The PureWick <sup>TM</sup> Urine Collection System is to be used with PureWick <sup>TM</sup> External Catheters which are intended for non- invasive urine output management. | <ul> <li>Discontinue use if an allergic reaction occurs. Not recommended for users who are experiencing skin irritation or skin breakdown in device contact areas.</li> <li>Keep small device parts, cords and tubing out of reach of children.</li> <li>Always unplug PureWick<sup>TM</sup> Urine Collection System</li> </ul> |


before cleaning or when not in use.

- DO NOT IMMERSE THE PUREWICK<sup>TM</sup> URINE COLLECTION SYSTEM IN WATER. As with most electrical devices, electrical parts in this system are electrically live even when the power is off. To reduce the risk of electric shock, if the PureWick<sup>TM</sup> Urine Collection System falls into water, unplug immediately. DO NOT REACH INTO THE WATER TO RETRIEVE IT.
- Do not use PureWick<sup>TM</sup> Urine Collection System in oxygen rich environments or in conjunction with flammable anesthetics.
- For PW200: The battery cells used in this device may present a fire or chemical hazard. To minimize the risk of damaging the battery inside the PureWick<sup>TM</sup> Urine Collection System, do not use the device outside the indicated operating temperature range of 41°F - 104°F (5°C -40°C). The battery is not intended to be replaced; replacement could result in a hazard.

# Study Intervention: Hollister® Female Urinary Pouch External Collection Device

Potential adverse events:

- Irritation
- Broken skin
- Rash
- Severe Redness
- Swelling

Hollister® Female Urinary
Pouch External Collection
Device is a urinary
collection pouch with a
skin barrier suitable for
frequent pouch changes or

To avoid potential adverse events, while using the Hollister® Female Urinary Pouch External Collection Device, it is advised


| • Itching or pain in vulva/perineal area | use on fragile skin. It is in | the product should not |
|---|---|---|
| • Fever | direct contact with the | reuse the pouch after |
| Abnormal Discharge | vulva or perineal area. | use. Reprocessing, cleaning, disinfection, and sterilization may comprise the product. • Urinary pouch should only be used under supervision of healthcare professional. • Urinary pouch should not be used on patients with any contraindications per IFU. |
| St | udy Procedures | |
| Potential loss of confidentiality of information | Study data, including photographs when applicable, will be collected in the home setting and transferred to the investigational site for collection in the clinical database. | Access controlled Secure File Transfer Protocol (SFTP) software will be used to transfer data to investigational site |

#### 2.5.1 Benefit Assessment

Potential benefits to participants using the PureWick<sup>TM</sup> System may include:

- The PureWick<sup>TM</sup> System can help make better sleep possible for women with incontinence and their caregivers.<sup>24</sup>
- The PureWick<sup>TM</sup> System may help reduce the need for multiple changes at night, or trips to the bathroom.
- The PureWick<sup>TM</sup> System is easy to set up, and the PureWick<sup>TM</sup> Female External Catheter can be placed in a few easy steps.
- PureWick<sup>TM</sup> FEC can decrease risk of moisture-associated skin damage compared to the use of absorbent products such as adult briefs, pads, or sheets.

Other potential benefits of study participation include:

- Participants receive enhanced follow up, including daily skin assessments and urine output management by a nurse.
- Participants contribute to the process of generating clinical evidence for urine output management solution in the home setting.
- Potential to benefit from future reimbursement of the PureWick system.


# 2.5.2 Overall Benefit: Risk Conclusion

Taking into consideration the measures to minimize risk to participants in this study, the potential risks identified in association with the PureWick<sup>TM</sup> System and the Hollister® Female Urinary Pouch External Collection Device are justified by the anticipated benefits that may be afforded to participants with urinary incontinence.

# 3.0 OBJECTIVES AND ENDPOINTS

| Objectives | Endpoints |
|---|---|
| Primary | |
| To compare efficacy and safety of PureWick <sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device | <ul> <li>Efficacy – Daily capture rate via bed pad weights and captured volume.</li> <li>Safety – Daily skin irritation score using the Draize Scale.</li> </ul> |
| Secondary | |
| To assess impact of PureWick <sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device on Nocturnal Incontinence related Quality of Life. | <ul> <li>Nocturia Quality of Life (N-QOL) score collected at baseline and every 2 weeks during treatment.</li> <li>PROMIS Sleep Disturbance score collected at baseline and every 7 days during treatment.</li> </ul> |
| Tolerability – To assess the tolerance of PureWick <sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device over the expected duration of use | Tolerability – Number of days of actual use of both devices & Discontinuation rate attributed to the device's inconvenience or discomfort |
| To assess participant device preference, comfort, and ease of use of PureWick <sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device To assess participant preference between the PureWick <sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device after study completion | <ul> <li>Overall comfort and ease of use scores on a 5-point Likert scale (brief questionnaire) collected at the end of each treatment phase.</li> <li>Overall preference via end of study participant preference survey administered at study completion</li> </ul> |
| Tertiary/Exploratory | |
| N/A | N/A |


#### 4.0 STUDY DESIGN

## 4.1 Overall Design

In this prospective, post-market, multi-site, open-label, crossover trial, women with urinary incontinence requiring the use of diapers (changes complets (Fr)) at night will be 1:1 randomized to a treatment sequence using two devices (PureWick<sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device) and followed for approximately 10 weeks through 2 treatment phases.

Approximately 30 female participants from 2 sites will be enrolled into the study. Those meeting eligibility criteria will be treated according to the treatment sequence assigned during randomization. Participants will be trained by the nurses for the applicable product at the beginning of each treatment phase and have access to the IFU to review during each treatment phase. The total expected duration of subject participation is approximately 10 weeks. Participants will use the device assigned in treatment phase 1 overnight while sleeping for 4 weeks (28 days) before transitioning to the second assigned device in treatment phase 2. There will be a minimum washout period of 2 weeks (not to exceed 4 weeks) between treatment phases and a re-screening of eligibility criteria before the second phase. Participants assigned to both treatment arms will place and remove the FEC (female external catheter) or FUP (Female Urinary Pouch) after standardized teaching is completed on the first day of the treatment phase.

The primary objectives are to evaluate safety (skin injury) and efficacy (capture rate). Safety will be assessed using the Draize Scale and efficacy will be measured based on daily urine capture rate. Nurses will visit participants' homes daily to perform a skin assessment and collect urine measurements during the treatment phases. Participants will be withdrawn from the treatment phase if grade 4 is achieved in any category on the Draize skin irritation scale.

The secondary objectives are to assess quality of life, tolerability, preference, comfort and ease of use. Quality of life will be measured using self-reported changes in quality of life via the validated Nocturia Quality of Life (N-QOL) and PROMIS Sleep Disturbance assessments. Preference, comfort and ease of use will be measured using subjective evaluations of the therapy via participant surveys. Tolerability will be measured by number of days of actual use of both devices, and discontinuation rate attributed to the device's discomfort or inconvenience.


## 4.2 Scientific Rationale for Study Design

This study will assess the performance of and user experience with PureWick<sup>TM</sup> System in a home setting. The endpoints chosen for the study were selected based on peer-reviewed research and feedback from expert consultants, Centers for Medicare & Medicaid Services, applicable health authorities and urology key opinion leaders.

To best mimic potential users of the PureWick™ System, participants ≥18 years of age will be enrolled with a target of at approximately 90% of participants ≥65 years of age. The treatment duration of 4 weeks for each investigational device was selected to allow sufficient time for a potential impact to quality of life. For this study, the baseline quality of life scores will be compared to mid-treatment scores and to post-treatment scores.

The PureWick<sup>TM</sup> System may provide improvements to urine output management, specifically in the home-setting. Additionally, the PureWick<sup>TM</sup> At-Home study is required to provide the needed information to properly execute a future global randomized control trial (RCT) with confidence of success.

### 4.3 Participant Input into Design

Not applicable.

## 4.4 End of Study Definition

A participant is considered to have completed the study after she has completed both treatment phases and all required questionnaires.

The end of the study is defined as the date of completion of the last participant in the study.

#### **5.0 STUDY POPULATION**

Adult female participants requiring urine output management overnight in the home setting will be recruited for this study by the study site from their current patient list. Study sites may advertise and recruit new patients if eligible participants from the patient list have been exhausted.

To best mimic potential users of the PureWick<sup>TM</sup> System, participants  $\ge$ 18 years of age will be enrolled. It is desired that at approximately 90% of participants are  $\ge$ 65 years of age. This study will enroll approximately 30 participants.


#### 5.1 Inclusion Criteria

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

- 1. Adult Female Participants ≥18 years of age at the time of signing the informed consent.
- 2. Currently use diapers or equivalent at night for urine capture ("Change complet" (FR))
- 3. Willing to comply with all study procedures in this protocol.
- 4. Provision of signed and dated informed consent form.

#### **5.2 Exclusion Criteria**

Participants are excluded from the study if any of the following criteria apply:

- 1. Has frequent episodes of bowel incontinence without a fecal management system in place; or
- 2. Has moderate to heavy menstruation and cannot use a tampon or menstrual cup; or
- 3. Has Urinary tract, vaginal or other chronic infections, active genital herpes; or
- 4. Has Urinary retention; or
- 5. Is agitated, combative, and/or uncooperative and may remove the external catheter or pouch; or
- 6. Has any wound, open lesion or irritation on the genitalia, perineum, or sacrum; or
- 7. Has any pre-existing neurological, psychiatric, or other condition that would confound quality of life assessment or would make it difficult to self-report on quality-of-life questionnaires in the opinion of the investigator; or
- 8. Is known to be pregnant at time of enrollment (for women of childbearing age); or
- 9. Any other condition that, in the opinion of the investigator, would preclude them from participating in the study.
- 10. Is under supervision of a legally authorized representative.

# 5.3 Lifestyle Considerations

No restrictions are required.

#### **5.4 Screen Failures**

Screen failures are defined as participants who consent to participate in the clinical study but do not subsequently meet eligibility criteria prior to treatment. Data collected for screen failures will include consent, randomization, criteria leading to exclusion, and AEs.

Individuals who do not meet the criteria for participation in this study (screen failure) may be rescreened if the exclusionary criteria are temporary in nature and may resolve over


time (e.g., active infection, open wound, etc.). Rescreened participants will receive a new

participant number.

### **6.0 STUDY INTERVENTION(S)**

## 6.1 Investigational/Test Device

The PureWick<sup>TM</sup> System includes the PureWick<sup>TM</sup> Female External Catheter and the PureWick<sup>TM</sup> Urine Collection System. The PureWick<sup>TM</sup> Female External Catheter (PureWick<sup>TM</sup> FEC) is marketed in both the United States and Europe. In the U.S. PureWick<sup>TM</sup> FEC is a Class I, 510(k) exempt device. In Europe, the PureWick<sup>TM</sup> FEC is a Class I, CE marked, non-sterile device.

The PureWick<sup>TM</sup> FEC is intended for non-invasive urine output management in female patients. The PureWick<sup>TM</sup> FEC (Figure 1) is a flexible, contoured external catheter that is positioned against the area where urine exits the female body. The PureWick<sup>TM</sup> FEC will be connected to the PureWick<sup>TM</sup> Urine Collection System (PUCS) via connector tubing. The PUCS uses suction (not felt by the user) to pull voided urine through the device. Urine continues through vinyl tubing until it reaches a collection canister, away from the body. The PureWick<sup>TM</sup> FEC and PUCS will be used according to the IFU.

# **6.2 Pre-placement Procedure**

Prior to placing the PureWick TM FEC, perineal care should be performed, and skin should be assessed for integrity.

Figure 1: PureWick<sup>TM</sup> Female External Catheter








Figure 2: PureWick<sup>TM</sup> Urine Collection System



All PureWick<sup>TM</sup> FECs and PUCS will be shipped directly to the study site from regular commercial stock. Access to the devices will be limited to study staff and will only be used by study participants who have provided written informed consent.

#### 6.3 Control Device/Standard of Care

The Hollister® Female Urinary Pouch External Collection Device will be used as a comparator for this study. The urinary collection pouch with a skin barrier is suitable for non-ambulatory females with urinary incontinence. It is designed to be emptied and should be attached to a drainage bag. The FUP is made with hydrocolloid skin adhesive and polymer/copolymer plastics.

## **6.4 Pre-placement Procedure**

To prepare the skin prior to placing the Hollister® FUP, the genital area should be washed with a mild soap and water and pubic hair trimmed. After drying the area thoroughly, the skin that will be in contact with the skin barrier may be wiped with a skin protective wipe if desired.

The pre-cut opening on the skin barrier can be modified so that it will encompass the urinary and vaginal orifices by cutting the opening with scissors.

If desired, barrier paste may be placed on the edge of the skin barrier that will adhere to areas where the skin surface is creased or uneven prior to placement.


Figure 3: Hollister® Female Urinary Pouch One-System and Bedside Drainage Bag



All Hollister® Female Urinary Pouch External Collection Devices will be shipped directly to the study site from regular commercial stock. Access to the devices will be limited to study staff and will only be used by study participants who have provided written informed consent.

# **6.5 Ancillary Devices/Products**

- PureWick<sup>TM</sup> replacement kit (PWKIT03) (US) and (PWKIT03E) (EU)
- Absorbent under-pads will be used to collect and measure urine leakage.
- Medium/Large sealing plastic bags
- Medical triangular graduated cylinders, 1000mL
- Commercially available scales will be used to weigh under-pads and mesh underwear. both before and after use to calculate urine capture rates.
- Bedside urine collection bags to capture outputs from the Hollister FUP
- Bedside urine bag holder
- Mesh Underwear
- PPE (gloves, chux)
- Barrier Paste
- Wipes
- Micropore tape
- Hair trimmers/clippers

## 6.6 Device Labeling

Commercial products will be supplied as labeled by the manufacturer. The test device and comparator products shall be labeled in accordance with regulatory requirements, including the following statement, "CAUTION - Investigational Device. Limited by Federal (or United States) law to investigational use." for the products used in the US, and with the following statement "exclusively for clinical investigation" for the devices used in France.


#### 6.7 Treatment Allocation and Measures to Minimize Bias

Known foreseeable factors that could potentially compromise the outcome of the investigation or interpretation of the results or introduce bias into the study are delineated in this section.

This is an open label, cross-over study in which each subject acts as her own control and therefore, the difference in treatments is derived from a within-subject comparison. This allows for better control of potential confounders and removes the inter-subject variability from the comparison between treatment groups. In addition, the study design includes a required washout period between treatment phases to minimize the impact of carry-over effect.

Standardized questionnaires and data collection tools will be used to assess participant preference and to document study findings, respectively. As training level and device experience could be a foreseeable factor that could impact study outcomes, standardized instructional videos will be used to train all participants on device use.

#### 6.8 Randomization

Subjects will be randomized 1:1 to the two sequences of treatment (using PureWick<sup>TM</sup> FECs in phase 1 and Hollister® Female External Pouch in phase 2, or the reversed order). This design allows the evaluation of elements such as the carryover effect, period effect, and sequence effect. To begin treatment phase in either the U.S. or France, using a prepared randomization schedule participants will be randomized 1:1 to use either PureWick<sup>TM</sup> FEC in phase 1 and Hollister® FUP in phase 2, or vice versa. Block randomization will be carried out using a fixed block size and stratified by investigational site and geography.

## 6.8.1 Blinding/Masking

Not applicable. This is an open-label study.

## **6.8.2** Procedures for Unblinding

Not applicable.

#### 7.0 STUDY PROCEDURES AND ASSESSMENTS

Study procedures and their timing are summarized in the Schema (Section 1.2). Protocol waivers or exemptions are not allowed. Adherence to the study design requirements, including those specified in the SoA, is essential and required for study conduct.


All screening evaluations must be completed and reviewed to confirm that potential participants meet all eligibility criteria. The investigator will maintain a screening log to record details of all participants screened and to confirm eligibility or record reasons for screening failure, as applicable.

# 7.2 Screening and Enrollment

#### 7.2.1 Informed Consent

The Principal Investigator or their designee will explain the study to the participant, answer all the participant's questions, and obtain written or electronic informed consent before the collection of any study data or performance of any study procedures in accordance with article 63 of the European Medical Device Regulations respectively CFR Parts 50 and 56 and any other applicable laws and regulations. The original copy of the consent will be retained with the participant records and a copy will be provided to the participant.

## 7.2.2 Eligibility

The participant's eligibility (inclusion/exclusion criteria) for study participation will be confirmed by the PI or designee (via on site or virtual visit (U.S. only)) per investigational site policy) and documented on the appropriate electronic case report form (eCRF). Participant baseline and demographic information, including, but not limited to age, sex assigned at birth, primary diagnosis, medical history, Katz ADL Index score and incontinence-specific information will be collected and recorded after informed consent is obtained prior to device use.

Participants who fail to meet eligibility criteria due to an exclusionary criterion that is temporary in nature and may resolve over time (e.g., active infection, open wound, etc.) can be rescreened at the PI's discretion.

### 7.2.3 Enrollment/ Assignment of Participant Number

Participants who sign an informed consent will be considered enrolled in this study.

A unique identification number will be given to study participants. Participant numbers will be assigned in sequential order. The participant number will consist of six digits. The first three digits will designate the site number and the last three digits will designate the participant number in sequential order.

#### 7.2.4 Randomization

Investigational sites will receive the randomization envelopes that are numbered in sequential orders. Within each randomization envelope, a treatment assignment card will be enclosed indicating which device to be used for each treatment phase. The

randomization envelope will be opened when all eligibility criteria are confirmed, and consent has been obtained. Randomization envelopes should be opened in sequential order. The treatment assignment card will be filed in the participant's record to serve as documentation. Participant randomization numbers will be captured in EDC.

#### 7.2.5 Home Nurse Introduction

The Principal Investigator or their designee will introduce enrolled participants to the nurse that will conduct daily home visits (either in person or virtually).

Nurse and participant will arrange the baseline visit. Once a baseline visit has been scheduled, the site coordinator/Pharmacist will reach out to Marken and setup study device shipment from clinical site to the Participant's home.

## 7.2.6 Day 1 - Baseline Assessments

This part of the study is to assess if the participants are eligible to begin treatment per assigned treatment schedule. During the baseline assessment urine output measurements will not be taken.

The nurse will collect nighttime routine (e.g., sleep position) and visually assess for any existing signs of irritation in the perineal area, using the Draize Scale Skin Scoring system.

#### If Skin Score is Greater than 0:

- 1. Participant is not eligible to begin treatment on that day.
- 2. Baseline visit can be rescheduled at the nurse's discretion within 2-4 weeks.
- 3. If the skin score of 0 is not achieved within 4 weeks from the original baseline visit, the participant will not be eligible for treatment.
- 4. Nurse will notify PI and Site staff will complete appropriate eCRFs.

## If Skin Score is 0:

- 1. Nurse will have participant complete Baseline N-QOL & PROMIS Sleep Disturbance assessment.
- 2. Nurse will confirm treatment assignment.
- 3. Nurse will provide device and procedure training via standardized product training video.
- 4. Once training is completed, nurse will ensure the participant have all the supplies prepped for the first night of device wear.
- 5. Nurse will pre-weigh and document weight of sealed bed pad in bag
- 6. If assigned to PureWick<sup>TM</sup> treatment phase, nurse will pre-weigh and document weight of canister before use.
- 7. If assigned to Hollister FUP treatment phase, nurse will pre-weigh and document weight of the graduated cylinder.
- 8. If applicable, nurse will pre-weigh and document weight of mesh underwear in bag.


9. Nurse will confirm next day visit with participant.

#### 7.2.7 Days 2-7

1. Prior to nurse visit, participants are expected to have placed the used night pads and mesh underwear (if applicable) in their respective labeled, pre-weighed sealed bag upon completion of sleep.

- 2. Nurse will weigh and document weight of night pads and mesh underwear (if applicable).
- 3. The nurse will weigh and document the captured urine.
  - For PureWick<sup>TM</sup> Treatment Phase the captured urine volume in the PW urine collection canister will be weighed and documented.
  - For Hollister® FUP Treatment Phase the captured urine volume in the bedside urine bag will be emptied into a graduated cylinder, then weighed and documented.
- 4. The nurse will note any signs of skin irritation or injury and document the Draize Scale score\*
- 5. If during the skin assessment a Draize score of 4 is documented on the skin irritation scale in any category, this must be recorded as an AE and will require participants to discontinue from the treatment phase; participant will immediately begin wash out period and complete N-QoL.
- 6. Nurse will pre-weigh and document weight of study supplies for next night use.
- 7. The nurse will confirm the next day visit.

#### \* For safety assessment, see section 7.3

#### 7.2.8 Day 8

- 1. Same procedures as days 2-7.
- 2. Participant to complete Day 8 PROMIS Sleep Disturbance assessment.

#### 7.2.9 Days 9-14

1. Same procedures as days 2-7.

#### 7.2.10 Day 15

- 1. Same procedures as days 2-7.
- 2. Participant to complete 2-week N-QOL assessment.
- 3. Participant to complete Day 15 PROMIS Sleep Disturbance assessment.

#### 7.2.11 Days 16-21

1. Same procedures as days 2-7.

#### 7.2.12 Day 22

- 1. Same procedures as days 2-7.
- 2. Participant to complete Day 22 PROMIS Sleep Disturbance assessment.


#### 7.2.13 Days 23-28

1. Same procedures as days 2-7.

## 7.2.14 Day 29

- 1. Same procedures as days 2-7 with the exception of steps 6 and 7.
- 2. Participant to complete 4-week N-QOL assessment.
- 3. Participant to complete Day 29 PROMIS Sleep Disturbance assessment.
- 4. Participant to complete comfort and ease of use questionnaires.
- 5. If this day is the last day of phase 1 treatment for the participant, they will begin washout and prepare for phase 2 treatment.
- 6. If this day is the last day of phase 2 treatment for the participant, they will complete the study. Participant is to complete the End of Study Preference Survey.

## 7.2.15 Day 30

The participant will be asked to report any discomfort or voiding issues occurring within the first 24 hours after treatment phase completion or discharge from the study to the PI or sponsor. Skin assessments will also be conducted 24 hours after the participant completes the treatment phase and/or the study.

## 7.2.16 Days 29-42 (+14) Wash Out Period

Participant begins washout period of 2 weeks (not to exceed 4 weeks) between treatment phase 1 and treatment phase 2. At the completion of washout, the nurse will perform a rescreening of eligibility criteria before phase 2 treatment begins.

#### 7.2.17 Treatment Phase 2

Same procedures as outline in sections 7.2 - 7.11.

#### 7.3 Safety Assessments

#### 7.3.1 Draize Scale

For each daily visit (described in 7.2-7.7), skin condition will be evaluated by nurses using the Draize scale (Table 1). Skin assessments will also be conducted 24 hours after the participant completes the study, either in person or virtually.

If during the skin assessment a Draize score of 4 is documented on the skin irritation scale in any category, it must be recorded as an AE and will require participants to discontinue from the treatment phase. Any other score on the skin irritation scale in any category may be recorded as an AE based on PI discretion.


To assess a potential AE identified during the home visit, the nurse will contact the PI or designee. The site will document the AE assessment on the appropriate CRF from and follow the AE until resolution. If the PI requests a follow up visit with the participant, this can be conducted on site or virtually per investigational site policy.

However, if the AE is not resolved during the treatment phase(s) within 4 weeks from the AE start date, the participant will be discontinued from the study.

Also, if during the skin assessment a Draize score of 2 or greater is documented for the device placement site, a <u>photograph may need to be taken of the skin in the anatomical area of device application.</u> The photo will be sent in a pseudonymized matter to the site, only the subject ID and the date when the picture was taken will be collected. These photographs will be shared with the Principal Investigator / Sub-Investigator, the Sponsor, and the study staff only and will be used for the Principal Investigator / Sub-Investigator 's review and assessment of the skin reactions.

Table 1: Draize Scale for Skin Irritation

| Score | Erythema (redness) | Edema (swelling) | Bleeding |
|---|---|---|---|
| 0 | None | None | None |
| <b>1</b> <sup>a</sup> | Very slight (barely perceptible) erythema | Very slight (barely perceptible) skin surface rise | Just a visible spot of red |
| 2ª | Well-defined erythema | Well-defined skin surface rise<br>(edges of area well-defined by<br>definite raising) | A drop of red blood |
| $3^a$ | Moderate erythema | Moderate skin surface rise | A continuing ooze of red blood |
| 4 <sup>b</sup> | Severe (beet red) or<br>damage to skin (eschar<br>formation) | Severe skin surface rise | Significant bleeding from the sight |

<sup>&</sup>lt;sup>a</sup> = Represents irritation in any category and may require participant's removal from the study based on PI decision

Note: a rating of 1-3 on the skin irritation scale in any category may be recorded as an AE based on PI discretion.

#### 7.4 User Preference Questionnaire

Prior to each treatment phase completion, the participant will be asked to complete a short questionnaire on their experience with the PureWick<sup>TM</sup> System or the Hollister® FUP. The questionnaire is designed to assess the following:

 $<sup>^{</sup>b}$  = A rating of 4 on the skin irritation scale in any category must be recorded as AE and will require participant's removal from the treatment phase and/or study.


• Comfort with PureWick<sup>TM</sup> FEC/PureWick<sup>TM</sup> Urine Collection System or the Hollister® Female Urinary Pouch External Collection Device

• Ease of use in placing and removing the PureWick<sup>TM</sup> FEC and the Hollister® Female Urinary Pouch External Collection Device

After completing both treatment phases for the study, the participant will complete the preference questions on their experience with the PureWick<sup>TM</sup> System and the Hollister® FUP. The survey is designed to assess the following:

• The participants preferred device after using both the PureWick<sup>TM</sup> FEC/PureWick<sup>TM</sup> Urine Collection System and the Hollister® Female Urinary Pouch External Collection Device.

## 7.5 Participant Follow-Up

After all procedures are complete in both treatment phases, the participant will be discharged from the study. The participant will be asked to report any discomfort or voiding issues occurring within the first 24 hours after discharge from the study to the PI or sponsor.

## 7.6 Replacement of Participants

A participant that discontinues from the study will be replaced when feasible.

#### 8.0 PARTICIPANT DISCONTINUATION/WITHDRAWAL

## 8.1 Discontinuation/Withdrawal

- A participant may withdraw from the study at any time at his/her own request or may be withdrawn at any time at the discretion of the investigator or sponsor for safety, behavioral, compliance, or administrative reasons. This is expected to be uncommon.
- At the time of discontinuing from the study, no further assessments will be performed.
- If the participant withdraws consent for disclosure of future information, the sponsor may retain and continue to use any data collected before such a withdrawal of consent.
- Participants who withdraw or discontinue the study early may be replaced.

#### 8.2 Lost to Follow-Up

A participant will be considered lost to follow-up if she repeatedly fails to keep the visit schedule or is unable to be contacted by the study site or nurses.

The following actions must be taken if a participant fails to keep the visit schedule or is unable to be contacted:


• The site and nurse must attempt to contact the participant and reschedule the missed visit as soon as possible and counsel the participant on the importance of maintaining the assigned visit schedule and ascertain whether or not the participant wishes to and/or should continue in the study.

- Before a participant is deemed lost to follow up, the investigator or designee must make every effort to regain contact with the participant. Where possible, 3 telephone calls and, if necessary, a certified letter to the participant's last known mailing address or local equivalent methods. These contact attempts should be documented in the participant's study record.
- Should the participant continue to be unreachable, she will be considered to have withdrawn from the study.

#### 9.0 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 9.1 Definitions of Events

#### 9.1.1 Adverse Events (AEs)

An AE is defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, users or other persons, whether or not related to the investigational device and whether anticipated or unanticipated (ISO14155:2020). This definition includes events related to the investigational device, the comparator or the procedures involved.

Pre-existing conditions should be considered as part of the participant's medical history and should not be reported as an AE unless there is a substantial increase in severity or frequency of the condition, which has not been attributed to natural history. Likewise, planned hospital visits and/or hospital stays should not be considered as adverse events. Exacerbation of an existing condition should be reported as an AE if the event meets the protocol definition of an AE.

The clinical course of the event will be followed according to accepted standards of medical practice until the event resolves, stabilizes, or in the opinion of the Investigator, is no longer considered clinically significant. The Investigator must supply the Sponsor with information concerning the follow up and/or resolution of the AE.

#### 9.1.2 Serious Adverse Events (SAEs)

A serious adverse event is defined by ISO 14155 and/or 21 CFR 803.3 as an adverse event that led to:

- a. Death.
- b. Serious deterioration in the health of the participant, users, or other persons as defined by one or more of the following:


• a life-threatening illness or injury, or

- a permanent impairment of a body structure or a body function including chronic diseases, or
- in-patient or prolonged hospitalization, or
- medical or surgical intervention to prevent life-threatening illness or injury, or permanent impairment to a body structure or a body function,
- c. Fetal distress, fetal death, a congenital abnormality, or birth defect including physical or mental impairment.

NOTE: Planned hospitalizations for a preexisting condition, or a procedure required by this trial without serious deterioration in health, is not considered an SAE.

## 9.1.3 Adverse Device Effect (ADE) / Serious Adverse Device Effect (SADE)

An adverse device effect is defined as any adverse event that is considered to be related to the use of an investigational medical device. This definition includes any event resulting from insufficiencies or inadequacies in the instructions for use, deployment, implantation, or operation or any malfunction of the investigational device and includes any event that is a result of a user error, intentional misuse of the investigational medical device and/or comparator if the comparator is a medical device.

A serious adverse device effect (SADE) is defined as an ADE that has resulted in any of the consequences characteristic of an SAE. An anticipated serious adverse device effect (ASADE) is an effect which by its nature, incidence, severity or outcome has been identified in the risk assessment.

#### 9.1.4 Unanticipated (Serious) Adverse Device Effect (UADE/USADE)

An unanticipated (serious) adverse device effect (UADE/USADE) is any (serious) adverse device effect on health or safety or any life-threatening problem or death caused by, or associated with, an investigational device, which by its nature, incidence, severity, or outcome has not been identified in the current instructions for use and/or current version of the risk analysis report, or any other unanticipated serious problem associated with a device that relates to the rights, safety or welfare of participants.

Anticipated serious adverse device effect (ASADE) is an effect which by its nature, incidence, severity or outcome has been identified in the risk assessment.

A sponsor shall immediately conduct an evaluation of any unanticipated adverse device effect.

UADEs/USADEs will be reported to FDA as required by 21 CFR Part 812 and ISO 14155:2020 and will be reported to the appropriate governing body per ISO 14155:2020.


## 9.2 Severity of Adverse Events

Each AE shall be assessed for its severity, or the intensity of an event, experienced by the participant according to the criteria below.

| Severity Rating | Description |
|---|---|
| Mild | Event, signs, or symptoms that do not interfere with the participant's daily activity, are usually considered self-limiting, can be treated with non-prescription type medications, and do not require medical intervention |
| Moderate | Event may interfere or cause low level inconvenience with the participant's daily activity. Requires medical intervention and/or treatment; however, unlikely to require hospitalization or be considered potentially life-threatening in nature |
| Severe | Event may cause significant discomfort to the participant and/or interferes with the participant's daily activity. Requires medical intervention and/or treatment to preclude a permanent impairment; may be life threatening and/or require hospitalization |

## 9.3 Relationship of Adverse Event to Device(s)/Procedure

Each AE will be assessed for its relationship to the investigational device or procedure according to the following guidelines.

- A. Assess each AE for its relationship to the device or procedure.
  - Device Related: This category should be restricted to AEs directly attributable to the PureWick<sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device during the urine capture assessments.
  - Procedure: A procedure includes any study-related activity performed during the set-up or application of the PureWick<sup>TM</sup> System and Hollister® Female Urinary Pouch External Collection Device and/or urine capture assessment procedure.
- B. To assess the causality, clinical judgement should be used and the relevant study documentation, such as the study protocol should be consulted. The presence of confounding factors, such as concomitant medication/treatment, underlying diseases, other concurrent illness or risk factors should also be considered. The above considerations apply also to the serious adverse events occurring in the comparison group.

Each SAE will be classified according to four different levels of causality:


1. Not Related

2. Possible

3. Probable

4. Causal Relationship

| Relatedness | Description |
|---|---|
| Not Related | Relationship to the device, comparator or procedures can be excluded when: • the event has no temporal relationship with the use of the investigational device, or the procedures related to application of the investigational device; • the serious adverse event does not follow a known response pattern to the medical device (if the response pattern is previously known) and is biologically implausible; • the discontinuation of medical device application or the reduction of the level of activation/exposure - when clinically feasible - and reintroduction of its use (or increase of the level of activation/exposure), do not impact on the serious adverse event; • the event involves a body-site or an organ that cannot be affected by the device or procedure; • the serious adverse event can be attributed to another cause (e.g. an underlying or concurrent illness/ clinical condition, an effect of another device, drug, treatment or other risk factors); • the event does not depend on a false result given by the investigational device used for diagnosis, when applicable; In order to establish the non-relatedness, not all the criteria listed above might be met at the same time, depending on the type of device/procedures and the serious adverse event. |
| Possible | The relationship with the use of the investigational device or comparator, or the relationship with procedures, is weak but cannot be ruled out completely. Alternative causes are also possible (e.g. an underlying or concurrent illness/ clinical condition or/and an effect of another device, drug or treatment). Cases where relatedness cannot be assessed, or no information has been obtained should also be classified as possible. |
| Probable | The relationship with the use of the investigational device or comparator, or the relationship with procedures, seems |


| 10 Арт 2024 | relevant and/or the event cannot be reasonably explained by |
|---|---|
| | another cause. |
| Causal<br>Relationship | the serious adverse event is associated with the investigational device, comparator or with procedures beyond reasonable doubt when: • the event is a known side effect of the product category the device belongs to or of similar devices and procedures; • the event has a temporal relationship with investigational device use/application or procedures; • the event involves a body-site or organ that • the investigational device or procedures are applied to; • the investigational device or procedures have an effect on; • the serious adverse event follows a known response pattern to the medical device (if the response pattern is previously known); • the discontinuation of medical device application (or reduction of the level of activation/exposure) and reintroduction of its use (or increase of the level of activation/exposure), impact on the serious adverse event (when clinically feasible); • other possible causes (e.g. an underlying or concurrent illness/ clinical condition or/and an effect of another device, drug or treatment) have been adequately ruled out; • harm to the subject is due to error in use; the event depends on a false result given by the investigational device used for diagnosis when applicable; In order to establish the relatedness, not all the criteria listed above might be met at the same time, depending on the type of device/procedures and the serious adverse event. |

## 9.4 Reporting of Events

For all adverse events, all sections of the appropriate electronic Case Report Form (eCRF) must be completed including AE start and end date, outcome of AE, severity, seriousness, relationship to device and relationship to the procedure. All AEs shall be promptly reported to the Sponsor.

For European site(s):

• All SAEs, SADEs, UADEs/USADEs, and Serious Health Threats must be reported to the Sponsor via completion of the appropriate eCRF no later than 3


calendar days of the site/investigator becoming aware of the event. If the study team is unable to access the electronic data capture system, the event may be reported to the Sponsor by emailing UCC.ClinicalSafety@bd.com.

• De-identified copies of all requested relevant documentation should be submitted to the Sponsor within 72 hours of knowledge, as appropriate.

#### For U.S. site(s):

- All SAEs, SADEs, UADEs/USADEs, and Serious Health Threats must be reported to the Sponsor via completion of the appropriate eCRF within 1 working day of the site/investigator becoming aware of the event. If the study team is unable to access the electronic data capture system, the event may be reported to the Sponsor by emailing UCC.ClinicalSafety@bd.com.
- De-identified copies of all requested relevant documentation should be submitted to the Sponsor within 72 hours of knowledge, as appropriate.

In the US, it is the responsibility of the Investigator to report adverse events to individual Institutional Review Boards (IRBs) and/or regulatory authorities according to the local regulations.

In Europe, it is the responsibility of the Sponsor to report adverse events to individual Ethics Committees (ECs) and/or regulatory authorities according to the local regulations in each participating country.

- For the purpose of this guidance and based on the definitions above, the following events are considered sponsor reportable events in accordance with MDR Art. 80(2):
  - a) any serious adverse event that has a causal relationship with the investigational device, the comparator or the investigation procedure or where such causal relationship is reasonably possible;
  - b) any device deficiency that might have led to a serious adverse event if appropriate action had not been taken, intervention had not occurred, or circumstances had been less fortunate;
  - c) any new findings in relation to any event referred to in points a) and b).

#### 9.5 Serious Health Threats

Serious Health Threats are a signal from any adverse event or device deficiency that indicates an imminent risk of death or a serious deterioration in the health in subjects, users or other persons, and that requires prompt remedial action for other subjects, users or other persons. This would include events that are of significant and unexpected nature such that they become alarming as a potential serious health hazard or possibility of multiple deaths occurring at short intervals (ISO14155:2020)


#### 9.6 Safety Committees

Not applicable.

#### 9.7 Device Deficiencies

The Investigator will record a device deficiency if a device used in the study procedure failed to meet its performance specifications in the identify, quality, durability, reliability, usability, safety or performance, including malfunction, use errors or in adequacy in information supplied by the manufacturer, mechanical failure, malfunction, or defect. Device deficiencies also include use errors and inadequate labeling. This applies to: devices used to treat the participant, or devices in which the package was opened, but the device was not used for treatment, or devices with which treatment was attempted, but the device did not remain through the entire study procedure/period.

All device deficiencies will be recorded on the appropriate Case Report Form and will be promptly reported to the Sponsor. All sections of the appropriate eCRF must be completed including date of deficiency, time of deficiency, device identifiers (i.e. lot number, serial number). The device(s) should be returned to the Sponsor as outlined in the site's regulatory binder.

If the device deficiency was associated with an AE, the reporting provisions for AEs, ADEs, SAEs, SADEs and UADEs/USADEs apply. If the device deficiency was not associated with an AE, an assessment of whether the device deficiency could have led to a SADE if suitable action had not been taken, if intervention had not been made or if circumstances had been less fortunate should be reported.

Reported deficiencies will be investigated and reported under 21 CFR part 803 Medical Device Reporting and ISO 14155:2020 by the Sponsor if necessary. The site may be contacted to provide additional information to allow the Sponsor to conduct a thorough investigation.

It is the responsibility of the Investigator for the U.S. and Sponsor for France to notify the IRB/EC of such device deficiencies in accordance with the IRB/EC and/or the Competent Authority's local regulations.

## 10.0 STATISTICAL METHODS

The statistical analysis plan will be finalized prior to database lock and will include a more technical and detailed description of the statistical analyses described in the following sections. Analyses will be performed per protocol and statistical analysis plan. Any deviation from planned analyses will be described in the clinical study report along with justification of change. This section includes a summary of the planned statistical analyses of the most important endpoints including primary and key secondary endpoints.


## 10.1 Overview of Study Design

This is a prospective, open-label, 2 by 2, crossover trial to evaluate the safety, efficacy, and patient quality of life of PureWick<sup>TM</sup> System in comparison with Hollister® Female Urinary Pouch. Participants are randomized 1:1 to use PureWick<sup>TM</sup> System in phase 1 and Hollister® Female External Pouch in phase 2, or to use Hollister® Female Urinary Pouch in phase 1 and PureWick<sup>TM</sup> System in phase 2. Each phase lasts 4 weeks, with a 2-4 week washout period between phase 1 and phase 2. Capture rates and Draize Scale are assessed daily during both phases. Quality of life is assessed at baseline and every 14 days during phases 1 and 2. User preference questionnaires are completed at the completion of each treatment phase. The primary efficacy endpoint is the mean of daily capture rate. The primary safety endpoint is the mean of daily assessments of Draize Scale.

## 10.2 Sample Size Considerations

Approximately 30 participants will be enrolled. The sample size is planned based on operational and practical considerations and is adequate for the purpose of this pilot study.

## **10.3** Analysis Population

The following populations are defined:

| Population | Description |
|---|---|
| Enrolled | Subjects who signed ICF. |
| Intent-to-Treat (ITT) | Subjects who signed ICF and randomized to a treatment |
| | sequence. |
| As-Treated (AT) | ITT subjects, grouped by actual treatment sequence, if different |
| | from planned treatment sequence. |
| Per-Protocol (PP) | ITT subjects without major protocol deviation. |

ITT population will be used for the analyses of endpoints. Sensitivity analyses may be carried out using AT or PP population.

#### **10.4 General Considerations**

#### 10.4.1 Handling of Missing Data

Endpoint data may be missing due to reasons including lost to follow-up or withdrawal of consent. Reason for missing endpoints will be reported. For the primary efficacy endpoint, if capture rate assessments are missing for part of a treatment phase, derivation of the primary efficacy endpoint will be based on


available data. For the primary safety endpoint, the main analysis will be based on evaluable data. Sensitivity analyses may be performed for the primary safety endpoint where missing data is imputed using methods including linear interpolation or last-observation-carry-forward.

## 10.4.2 Poolability of Data

The effect of investigational site will be evaluated using regression models, with primary endpoint as the dependent variable, and treatment, investigational site, and the interaction term between treatment and investigational site as fixed effects.

#### 10.4.3 Multiplicity Control

No formal hypothesis test is planned for this pilot study. P values and confidence intervals may be provided for exploratory purposes and are unadjusted for multiplicity.

#### 10.5 Primary Endpoint(s)

## **10.5.1 Primary Efficacy Endpoint**

Capture rates is evaluated daily during participant phase 1 and phase 2. Daily capture rate is defined as:

captured urine weight / (captured urine weight + leaked urine weight)

The primary efficacy endpoint is derived by computing the mean of daily capture rate during each phase. Descriptive statistics of the primary efficacy endpoint, including mean, standard deviation, median, and range will be provided by treatment. The paired difference in mean daily capture rate between treatments will be provided.

#### 10.5.2 Primary Safety Endpoint

The primary safety endpoint is derived by computing the mean of Draize Scale assessed daily during each phase. Descriptive statistics of the primary safety endpoint, including mean, standard deviation, median, and range will be provided by treatment. Paired difference in mean daily Draize Scale between treatment will be provided.

## 10.6 Secondary Endpoint(s)

## 10.6.1 Questionnaire Nocturia Quality of Life (N-QoL)

The questionnaire consists of 13 items with a total score ranging from 0 to 52 higher score indicating greater impact of nocturia on quality of life). Descriptive statistics will be provided by treatment and by visit. Mixed effect linear regression model may be used, with treatment and sequence as the fixed effect, and participant as the random effect.


## 10.6.2 Questionnaire PROMIS Sleep Disturbance

Items in the questionnaire will be summarized both as categorical variable (using frequency count and percentage) and as continuous variables (using mean, standard deviation, median, and range) by treatment.

#### 10.6.3 Tolerability - Number of days of actual use

Number of days of actual use will be summarized using descriptive statistics by treatment. Paired difference between treatment will be provided.

#### 10.6.4 Tolerability - Discontinuation rate due to device discomfort or inconvenience

Rate of not completing a treatment phase due to device discomfort or inconvenience will be summarized using descriptive statistics.

## 10.6.5 Comfort, Ease of Use and Confidence

Items in the questionnaire will be summarized both as categorical variable (using frequency count and percentage) and as continuous variables (using mean, standard deviation, median, and range) by treatment.

#### 10.7 Tertiary/Exploratory Endpoint(s)

Not applicable.

#### 10.8 Other Analyses

Not applicable.

#### 10.9 Interim Analyses

Not applicable.

#### 11.0 DATA COLLECTION AND RECORD MAINTENANCE

#### 11.1 Case Report Forms

The Investigator is responsible for ensuring the completeness and accuracy of all study documentation.

All required clinical data will be collected/documented in sponsor-provided web-based electronic Case Report Forms (eCRFs). The eCRFs are designed to accommodate the specific elements of this clinical investigation and it is the responsibility of the Investigator to confirm that the data is completely and accurately entered in the appropriate sections of


the eCRF. Data reported on the eCRFs shall be derived from, and be consistent with, source documents and will be approved by the Investigator. An audit trail of changes or corrections to eCRFs will be maintained. Discrepancies between the source documents and the eCRFs shall be explained in writing. FDA 21 CFR 11 and ISO 14155:2020, 7.8.3 are followed as well as other applicable legislation on the handling of electronic data. Modification of the CRFs will only be made if deemed necessary by the Sponsor and/or the appropriate regulatory body.

Site numbers and Participant numbers will be used to track participant information throughout the study. Participant personal information will be de-identified.

#### 11.2 Source Documentation

Original or certified copies of all relevant clinical findings, observations, and other activities throughout the clinical investigation must be recorded and maintained in the study file of each enrolled participant.

## 11.3 Data Management

Data management is the responsibility of the Sponsor. Data from completed CRFs will be managed in a secured, controlled database. A Data Management Plan (DMP) will be developed that outlines the procedures used for database design and testing, database security, data review, database cleaning and issuing/resolving data queries. Procedures for validations, database finalization and data storage will also be contained within the DMP. Observation data will be collected prospectively at the time of each urine output monitoring event. As such, any missing data or inconsistent data cannot be retrieved from an alternate source. Particular care must be taken to ensure that all data are recorded in a clear and complete manner.

#### 11.4 Record Retention

For United States: The Investigator shall retain all study records for a minimum of two (2) years after the later of the following two dates: the date on which the study is terminated/completed or the date that the records are no longer required for purposes of supporting a pre-market approval application or a notice of completion of a product development protocol (21 CFR Part 812.140). The data for some of these records may be available in computerized form but the final responsibility for maintaining study records remains with the Investigator.

For European sites: Documentation shall be kept for a period of at least 10 years after the clinical investigation with the device in question has ended, or, in the event that the device is subsequently placed on the market, at least 10 years after the last device has been placed on the market.

The Investigator may withdraw from the responsibility to maintain records for the period required by transferring custody of the records to any other person who will accept responsibility for retaining them. Notice of a transfer shall be given to the Sponsor and


FDA, if applicable, not later than ten (10) working days after the transfer occurs.

## 12.0 QUALITY CONTROL AND ASSURANCE

## 12.1 Control of Study Products

Investigational study products will be released only for use by Investigators who have obtained written IRB/EC approval (as required) for participation in this study, who have completed all required study documentation, and who have been qualified by the Sponsor. Investigators must maintain control over all study products, and ensure they are used in accordance with this protocol. Failure to do so may result in the Sponsor suspending or terminating the study at the Investigator's site.

The Investigator will ensure that study products are only dispensed to participants (or used for specimens) properly enrolled in the study. The Investigator must maintain records of receipt, disposition, return and/or destruction of all study products. All investigational study products released to the site must be accounted for at the unit level prior to study close out, regardless of disposition. The Sponsor-Monitor will regularly review all records regarding study product accountability.

The Sponsor will maintain records that document the shipment, receipt, disposition, return and/or destruction of study products. A Study Supply Plan will be developed that contains study material traceability information and labeling requirements. Study product handling and accountability procedures will be outlined in the Clinical Monitoring Plan (CMP).

## 12.2 Monitoring

The Sponsor will designate trained and qualified personnel to monitor the progress of this clinical study in accordance with established standard operating procedures and the study-specific Monitoring Plan.

Prior to study start, a site initiation visit (SIV) will be conducted to review with the Investigator(s) and staff the provisions and proper conduct of this study. This visit will include a detailed review of this protocol, verification that all necessary documents are on file at the investigational site and confirmation of IRB/EC approvals.

During the study, routine monitoring visits (RMVs) will be conducted to assure the site continues to adhere to the protocol, the investigator agreement, and regulations regarding conduct of clinical studies. The Sponsor-Monitor will confirm that the ICF to be used is the version approved by the IRB/EC, confirm the applicable national privacy laws have been followed, verify that all necessary documents are on file at the investigational site and confirm that there are provisions to continue and maintain all documents and records throughout the study as required by applicable regulations. These monitoring visits will assess continued protocol compliance, adequate participant enrollment, accurate data reporting, monitoring of participant safety through identification and/or review of any device-related AEs, UADEs, or SAEs, device accountability, continued maintenance and


calibration of study-specific equipment (if applicable), and continued IRB/EC acceptance of the study.

At the completion of the study, the Sponsor-Monitor will conduct a final close-out visit or COV. The purpose of this visit may include but is not limited to collecting all outstanding study data documents, confirming that the Investigator's files are accurate and complete, reviewing the record retention requirements with the Investigator, providing for the return of unused devices to the Sponsor, reviewing records which account for device shipments and ensuring that all applicable requirements for closure of the study are met.

## 12.3 Audits and Inspections

If the study is selected for audit by the Sponsor or if there is an inspection by the appropriate Health Authorities, the Investigator and his team will make themselves available during the visit. The Investigator must agree to the inspection of all study related records and give the auditor/inspector direct access to source documents for verification of data on CRFs. The participant's anonymity must be ensured, and data checked during the audit must remain confidential.

As soon as the Investigator is aware of an upcoming inspection/audit by the Health Authorities, he/she will promptly inform the Sponsor. As agreed with the Investigator, Sponsor personnel may be present at the site during the inspection.

#### **12.4 Protocol Deviations**

A protocol deviation is defined as an event where the Investigator or site personnel did not conduct the study according to the protocol.

Except when necessary to protect the life or physical well-being of a participant, protocol deviations are not permitted. The Sponsor and the investigational site's IRB/EC must be notified immediately if an emergency situation arises in which the safety of a participant may require immediate intervention different than that defined in the protocol. This must be followed by written confirmation that describes the emergency action and outcomes, within five (5) working days from the date of the emergency action in accordance with the governing IRB/EC's requirement.

It is the Investigator's responsibility to ensure that there are no deviations from the Protocol. Except in an emergency, when a protocol deviation is planned or anticipated, the Sponsor should be contacted for approval. Any and all deviations must be recorded on the appropriate CRF regardless of whether medically justifiable or sponsor approved. Upon evaluation by the Sponsor, actions may be required to prevent additional deviations, such as retraining of the site, implementation of additional site procedures, and more frequent monitoring. If these steps fail, more serious measures, up to and including termination of enrollment at the site.


## 13.0 ADMINISTRATIVE REQUIREMENTS

### 13.1 Investigator and Site Selection

The Investigator must be of good standing as an Investigator and knowledgeable in relevant areas of clinical research to ensure adherence to the requirements of this protocol, including the protection of human participants. Other site personnel must have appropriate research experience and infrastructure to ensure adherence to this protocol and enrollment of sufficient numbers of evaluable participants. The curriculum vitae (CV) of the Investigator(s), Sub-Investigator(s) and Study Coordinator(s) will be maintained in the Sponsor's files as documentation of qualification by training and experience.

The Principal Investigator will sign the Investigator Agreement pages of this protocol, agreeing to comply with all applicable regulations and the requirements of this study as per the clinical study agreement. Federal databases will be searched to ensure that the Investigator(s) and/or the site are not prohibited from engaging in federally sponsored clinical research.

Any site that is deactivated prior to initial enrollment, either by the Sponsor or by the individual site itself, may be replaced.

## 13.2 Training

In addition to each Investigator and appropriate site personnel being trained on this protocol and study procedures during the Site Initiation Visit, product training will be provided by the Sponsor or designee and is required for each Investigator. Additional study staff (e.g., Sub-Investigator(s)) will also require device training provided from the Sponsor or proctoring by the PI. All training will be documented and filed at the investigational site and with the Sponsor.

## **13.3 Required Documents**

An Investigator may not screen or enroll participants until authorized to do so by the Sponsor. At a minimum, the following documentation should be received by the Sponsor prior to the commencement of study activities:

- Fully executed Non-disclosure Agreement (NDA) between PI/site and Sponsor;
- CVs, signed and dated within 2 years of study start for the PI and Sub-Investigator(s);
- CVs for Study Coordinator(s);
- Signed CSA by PI/site (or designee);
- Signed Investigator Agreement Page by PI and Sub-Investigator(s);
- Signed Financial Disclosure Statement by PI and Sub-Investigator(s);
- Completed and Signed Training Log by PI and Sub-Investigator(s);
- Study Personnel Identification list;
- Written approval from the IRB/EC of both the protocol and ICF, and any other applicable protocol specific material; and


• IRB/EC Membership List, Assurance of Compliance Form (for US only), or equivalent.

## 13.4 Publication Policy

The sponsor believes that results of applicable clinical studies should be published in peer-reviewed literature in a timely, accurate, complete and balanced manner, regardless of study outcomes, whenever possible. As such, at the conclusion of this study, an article may be prepared for publication in a reputable scientific journal. Formal presentation(s) or publication(s) of data collected from this study will be considered as a joint publication by the investigator(s) and the appropriate personnel of the Sponsor. Authorship will be based on generally accepted criteria of the ICMJE (International Committee of Medical Journal Editors) and determined by mutual agreement.

The publication of the principal results from any single-center experience within the study is not allowed until the preparation and publication of the multicenter results. Exceptions to this rule require the prior approval of the Sponsor. The analysis of other pre-specified and non-pre-specified endpoints will be performed by the Sponsor or its designee. Such analyses, as well as other proposed investigations or manuscripts will require the approval of the Sponsor.

#### 13.5 Study Registration

In compliance with Title VIII of Public Law 110-85, known as FDA Amendments Act of 2007 (FDAAA), the Sponsor will register this study studies and disclose study results in a publicly accessible database (i.e., ClinicalTrials.gov). This study will be registered no later than 21 days after commencing enrollment. Study results will be posted to the website within 12 months of the last participant visit for collection of primary outcome data.

In accordance with the Declaration of Helsinki, a description of the clinical investigation will be registered in a publicly accessible database before the start of recruitment activities and the content shall be updated throughout the conduct of the clinical investigation and the results entered at completion of the clinical investigation (ISO14155:2020).

#### 13.6 Termination of Study

The Sponsor reserves the right to suspend enrollment or terminate the study at any time for any reason. The Sponsor may suspend enrollment or terminate the study at a specific investigational site for reasons including, but not limited to, inadequate data collection, low participant enrollment rate, achievement of the total enrollment, conditions imposed by the reviewing IRB/EC and/or non-compliance with this protocol or other clinical research requirements. Written notice will be submitted to the Investigator in advance of such termination.

In the event of study suspension or termination, the Sponsor will send a report outlining the circumstances to the IRB/EC, and all Investigators and Regulatory Authorities as


required by regulation. If the study was terminated, resumption would be done according to 21 CFR Part 812.

#### 14.0 ETHICAL AND REGULATORY CONSIDERATIONS

#### 14.1 IRB/EC Approval

Investigators or designees must submit the study protocol, Informed Consent Form (if applicable), and all other locally required documentation to an appropriate IRB/EC and obtain study-specific written approval (favorable opinion) before being allowed to participate in the study. Before commencement of the study, the Investigator or designee must provide the Sponsor with written documentation of such approval. If applicable, the IRB/EC must give written renewal of the original approval at least annually to continue the study. A copy of the written renewal must be provided to the Sponsor.

The IRB/EC will be notified of any amendments to the protocol, as well as possible associated information and consent form changes, where applicable, and written approval (favorable opinion) will be obtained prior to implementation, as applicable.

The Investigator or designee is responsible for fulfilling any conditions of approval imposed by the IRB/EC, such as regular safety reporting, study timing, etc. The Investigator or designee will provide the Sponsor with copies of such reports.

## 14.2 Informed Consent and Confidentiality

Prior to any study procedure, the Investigator (or designee) must explain to each participant in layman's terms, the nature of the study, its purpose, expected duration, and the risks and benefits of study participation. Also, participant will be informed of uses and disclosures of their medical information for research purposes, and their rights to access information about them. All applicable national privacy laws (e.g., HIPAA requirements in the U.S., General Data Protection Regulation [GDPR] requirements in the EU) will be followed in this study. The participants must be informed of their right to withdraw from the study at any time and for any reason without sanction, penalty, or loss of benefits to which they are otherwise entitled, and that withdrawal from the study will not jeopardize their future medical care. Participants will be informed of their right to new information and/or findings relating to the clinical study, and the process by which this information is made available. After this explanation, given sufficient time to decide whether to participate, before any study procedure is conducted, and before entering the study, the participant must voluntarily provide consent in accordance with 21 CFR Parts 50 and 56 and ISO 14155:2020(E). The participant will receive a copy of his/her signed ICF.


## 14.3 Confidentiality

Participant confidentiality must be strictly held in trust by the Investigator, study staff, and the Sponsor. Participant confidentiality and anonymity will be maintained by removal of identifiers from any data, documentation, or clinical samples submitted to the Sponsor.

Any data collected meeting the definition of protected/confidential health information or personal identifying information will be collected and maintained using the designated authorizations and following privacy procedures as specified in the applicable health authority regulations.

The Sponsor-Monitor, authorized representatives of the sponsor, and/or applicable Health Authorities may inspect all documents and records required to be maintained by the Investigator. The Investigator/Site will permit access to such records.

#### 14.4 Regulatory Status

The PureWick<sup>TM</sup> System, comprised of the PureWick<sup>TM</sup> Female External Catheter and the PureWick<sup>TM</sup> Urine Collection System, is a Class I, 510(k) exempt device currently marketed in the United States and will be evaluated for its approved indication. The investigational device is CE marked and will be studied in a post-market fashion in Europe.

The Sponsor has determined this to be a non-significant risk study. Institutional Review Board (IRB) or Ethics Committee (EC) submission of this study plan along with IRB/EC study approval or waiver is required. The study will comply with the abbreviated IDE requirements under CFR 812.2 (b).

#### 14.5 Statement of Compliance

This clinical investigation will be conducted in compliance with the investigator agreement, protocol and following regulatory requirements:

- 21 CFR 50, 54, 56 and 812;
- 21 CFR 812 (Good Clinical Practice);
- ISO14155:2020 (Good Clinical Practice);
- EU MDR (Council Regulation 2017/745 of 5 April 2017)
- MDCG guidelines
- Ethical principles that have their origin in the Declaration of Helsinki; and
- Applicable sections of the national laws and regulations.

The clinical investigation will not commence at a clinical site until approval (favorable opinion) from the respective IRB/EC has been received. All additional requirements imposed by the IRB/EC(s) will be followed. Involvement of the national competent authorities (e.g. by notification, seeking authorization) will be accomplished as required by national laws and regulations.


#### 15.0 REFERENCES

- 1. Sørbye, L. W., Finne-Soveri, H., Ljunggren, G., Topinkova, E., Garms-Homolova, V., Jensdóttir, A. B., ... & AdHOC Project Research Group. (2009). Urinary incontinence and use of pads—clinical features and need for help in home care at 11 sites in Europe. Scandinavian journal of caring sciences, 23(1), 33-44.
- 2. Drennan, V. M., Cole, L., & Iliffe, S. (2011). A taboo within a stigma? A qualitative study of managing incontinence with people with dementia living at home. *BMC* geriatrics, 11(1), 1-7.
- 3. Drennan, V. M., Greenwood, N., Cole, L., Fader, M., Grant, R., Rait, G., & Iliffe, S. (2012). Conservative interventions for incontinence in people with dementia or cognitive impairment, living at home: a systematic review. *Bmc Geriatrics*, 12(1), 1-10.
- 4. Beer, J. M., McBride, S. E., Mitzner, T. L., & Rogers, W. A. (2014). Understanding challenges in the front lines of home health care: a human-systems approach. *Applied Ergonomics*, 45(6), 1687-1699.
- 5. Kuil, S. D., Hidad, S., Fischer, J. C., Visser, C. E., van Leth, F., de Jong, M. D., & Schneeberger, C. (2021). Diapers as Promising Alternative Collection Method for Urine Specimens in Nursing Home Residents: A Noninferiority Study. *Journal of the American Medical Directors Association*, 22(6), 1222-1227.
- 6. Hawkins, K., Pernarelli, J., Ozminkowski, R. J., Bai, M., Gaston, S. J., Hommer, C., ... & Yeh, C. S. (2011). The prevalence of urinary incontinence and its burden on the quality of life among older adults with medicare supplement insurance. *Quality of life research*, 20(5), 723-732.
- 7. Li, Y., Cai, X., Glance, L. G., & Mukamel, D. B. (2007). Gender differences in healthcare-seeking behavior for urinary incontinence and the impact of socioeconomic status: a study of the Medicare managed care population. *Medical care*, 1116-1122.
- 8. Mardon, R. E., Halim, S., Pawlson, L. G., & Haffer, S. C. (2006). Management of urinary incontinence in Medicare managed care beneficiaries: results from the 2004 Medicare Health Outcomes Survey. Archives of internal medicine, 166(10), 1128-1133.
- 9. Samuelsson, E., Victor, A., & Tibblin, G. (1997). A population study of urinary incontinence and nocturia among women aged 20-59 years. Acta obstetricia et gynecologica Scandinavica, 76(1), 74-80.
- 10. Bresee, C., Dubina, E. D., Khan, A. A., Sevilla, C., Grant, D., Eilber, K. S., & Anger, J. T. (2014). Prevalence and correlates of urinary incontinence among older, community-dwelling women. *Female pelvic medicine & reconstructive surgery*, 20(6), 328.
- 11. Goode PS, Burgio KL, Redden DT, et al. Population based study of incidence and predictors of urinary incontinence in black and white older adults. J Urol. 2008;179:1449–1453. discussion 1453–1444.
- 12. Beeckman, D. (2017). A decade of research on incontinence-associated dermatitis (IAD): evidence, knowledge gaps and next steps. *Journal of tissue viability*, 26(1), 47-56.
- 13. Coyne, K. S., Wein, A., Nicholson, S., Kvasz, M., Chen, C. I., & Milsom, I. (2014). Economic burden of urgency urinary incontinence in the United States: a systematic review. Journal of Managed Care Pharmacy, 20(2), 130-140.


- 14. Dramé, M., Fierobe, F., Lang, P. O., Jolly, D., Boyer, F., Mahmoudi, R., ... & Novella, J. L. (2011). Predictors of institution admission in the year following acute hospitalisation of elderly people. The journal of nutrition, health & aging, 15(5), 399-403.
- 15. Sura, S., Shiozawa, A., Ng, D., & Aparasu, R. R. (2021). Higher resource utilization and costs in long-term nursing home residents with overactive bladder: a retrospective study of medicare beneficiaries. Journal of the American Medical Directors Association, 22(6), 1300-1306.
- 16. T.W. Hu, T.H. Wagner, J.D. Bentkover, et al. Costs of urinary incontinence and overactive bladder in the United States: A comparative study. Urology, 63 (2004), pp. 461-465
- 17. M.L. Ganz, A.M. Smalarz, T.L. Krupski, et al. Economic costs of overactive bladder in the United States. Urology, 75 (2010), pp. 526-532.e1–18
- 18. A. Yehoshua, M. Chancellor, S. Vasavada, et al.
- 19. Health resource utilization and cost for patients with incontinent overactive bladder treated with anticholinergies. J Manag Care Spec Pharm, 22 (2016), pp. 406-413
- 20. E.O. Caplan, I.M. Abbass, B.T. Suehs, et al. Impact of coexisting overactive bladder in medicare patients with osteoporosis. Arch Gerontol Geriatr, 75 (2018), pp. 44-50
- 21. E. Durden, D. Walker, S. Gray, et al. The direct and indirect costs associated with overactive bladder within a commercially-insured population in the United States. J Occup Environ Med, 60 (2018), pp. 847-852
- 22. E. Durden, D. Walker, S. Gray, et al. The economic burden of overactive bladder (OAB) and its effects on the costs associated with other chronic, age-related comorbidities in the United States. Neurourol Urodyn, 37 (2018), pp. 1641-1649
- 23. Welk, B., & Kennelly, M. (2022). The relative importance of different consequences of nocturnal enuresis among older women: A conjoint analysis experiment. Neurourology and Urodynamics, 41(6), 1451-1457.
- 24. Khosla, L., Sani, J. M., & Chughtai, B. (2022). Patient and caretaker satisfaction with the PureWick system. The Canadian Journal of Urology, 29(4), 11216-11223.
- 25. Abraham, L., Hareendran, A., Mills, I. W., Martin, M. L., Abrams, P., Drake, M. J., ... & Noble, J. G. (2004). Development and validation of a quality-of-life measure for men with nocturia. *Urology*, 63(3), 481-486.
- 26. Mock, L. L., Parmelee, P. A., Kutner, N., Scott, J., & Johnson II, T. M. (2008). Content validation of symptom-specific nocturia quality-of-life instrument developed in men: issues expressed by women, as well as men. *Urology*, 72(4), 736-742.
- 27. Takao, T., Tsujimura, A., Kiuchi, H., Takezawa, K., Okuda, H., Yamamoto, K., ... & Nonomura, N. (2013). Correlation between overactive bladder symptoms and quality of life in Japanese male patients: focus on nocturia. *Urology*, 82(1), 189-193.
- 28. Incontinence urinaire. (n.d.-b). Urofrance. <a href="https://www.urofrance.org/patient/pathologies-urologiques/incontinence-urinaire/">https://www.urofrance.org/patient/pathologies-urologiques/incontinence-urinaire/</a>
- 29. Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID: 20685078; PMCID: PMC2965562.


#### 16.0 APPENDICES

## **Appendix 1: Draize Scale for Skin Irritation**

#### **Draize Scale for Skin Irritation**

| Score | Erythema (redness) | Edema (swelling) | Bleeding |
|---|---|---|---|
| 0 | None | None | None |
| 1 | Very slight (barely perceptible) erythema | Very slight (barely perceptible) skin surface rise | Just a visible spot of red |
| 2 | Well-defined erythema | Well-defined skin surface rise<br>(edges of area well-defined by<br>definite raising) | A drop of red blood |
| 3 | Moderate erythema | Moderate skin surface rise | A continuing ooze of red blood |
| 4 | Severe (beet red) or<br>damage to skin (eschar<br>formation) | Severe skin surface rise | Significant bleeding from the sight |

Reference: Draize J.H., Woodward G., Calvery H.O. Method for the study of irritation and toxicity of substances applied topically to the skin and mucous membranes. *J Pharmacol Exp Ther.* 1944; 82: 377-390

## **Appendix 2: Katz ADL assessment Score**

Appendix 3: PureWick<sup>TM</sup> Female External Catheter Instructions for Use PWFX30 (US)

Appendix 4: PureWick<sup>TM</sup> Female External Catheter Instructions for Use PWFX30E (EU)

Appendix 5: PureWick™ Urine Collection System Instructions for Use PW100 & PW 200 (US)

Appendix 6: PureWick™ Urine Collection System Instructions for Use PW200E (EU)

**Appendix 7: Hollister® Female Urinary Pouch External Collection Device Instructions for Use** 


Appendix 8: N-QOL English

Appendix 9: N-QOL French

**Appendix 10: PROMIS English** 

**Appendix 11: PROMIS French** 

Appendix 12 : Participant Comfort Questionnaire PureWick™ System (Sample)

| Participant Number: | | Visit#: | | |
|---|---|---|---|---|
| Now that you have experienced the use of each device as well as voiding with the device in place, please answer the following questions. | | | | |
| 1. On a scale of 1 to 5 where 1 is very uncomfortable and 5 is very comfortable, how comfortable was the <u>placement</u> of the PureWick <sup>TM</sup> Female External Catheter? | | | | |
| 1 | 2 | 3 | 4 | 5 |
| Very<br>uncomfortable | Uncomfortable | Neither comfortable nor uncomfortable | Comfortable | Very<br>Comfortable |
| Comments: | | | | |
| | to 5 where 1 is very<br>ne PureWick <sup>TM</sup> Syst | uncomfortable and<br>em during sleep? | 5 is very comfortab | le, how |
| 1 | 2 | 3 | 4 | 5 |
| Very | Uncomfortable | Neither | Comfortable | Very |
| uncomfortable | | comfortable nor uncomfortable | | Comfortable |
| Comments: | | | | |
| | | uncomfortable and reWick <sup>TM</sup> Female F | | le, how |
| 1 | 2 | 3 | 4 | 5 |
| Very<br>uncomfortable | Uncomfortable | Neither comfortable nor uncomfortable | Comfortable | Very<br>Comfortable |
| Comments: | | | | |


| 2 a.c. 10 11p1 202 . | | | | |
|---|---|---|---|---|
| 4. On a scale of 1 | to 5 where 1 is very | unlikely and 5 is ve | ery likely, how likel | v would you be to |
| | - | o one of your loved | • | J J |
| | ife wick bystem to | o one of your loved | ones: | |
| 1 | 2 | 3 | 4 | 5 |
| Very unlikely | Unlikely | Neither likely | Likely | Very Likely |
| | | nor unlikely | | |
| Comments: | | | | |

# Appendix 13 : Participant Comfort Questionnaire Hollister® Female Urinary Pouch External Collection Device (Sample)

| Participant Number: | | | Visit#: | |
|---|---|---|---|---|
| <del>-</del> | Now that you have experienced the use of each device as well as voiding with the device in place, please answer the following questions. | | | |
| | • | | d 5 is very comfortab<br>Urinary Pouch Exter | |
| 1 | 2 | 3 | 4 | 5 |
| Very<br>uncomfortable | Uncomfortable | Neither comfortable nor uncomfortable | Comfortable | Very<br>Comfortable |
| Comments: | | | | |
| 2. On a scale of 1 to 5 where 1 is very uncomfortable and 5 is very comfortable, how comfortable was the Hollister® Female Urinary Pouch External Collection Device during sleep? | | | | |
| 1 | 2 | 2 3 4 5 | | |
| Very Uncomfortable Very uncomfortable Uncomfortable Very uncomfortable Comfortable Comfortable Comfortable | | | | |


| Comments: | | | | |
|---|---|---|---|---|
| 2 0 | 4-5-11: | | 5: | 1. 1 |
| | | | 5 is very comfortabinary Pouch Externa | |
| Device? | | | | |
| 1 | 2 | 3 | 4 | 5 |
| Very | Uncomfortable | Neither | Comfortable | Very |
| uncomfortable | | comfortable nor uncomfortable | | Comfortable |
| Comments: | | | | |
| | | - | ery likely, how likel | |
| | ollister® Female Ur | inary Pouch Externa | al Collection Device | to one of your |
| loved ones? | loved ones? | | | |
| 1 | 2 | 3 | 4 | 5 |
| Very unlikely | Unlikely | Neither likely nor unlikely | Likely | Very Likely |
| Comments: | | | | |

## Appendix 14: PureWick<sup>TM</sup> System Participant Ease of Use Questionnaire (Sample)

| Participant Number: | | V1S1t #: | | |
|---|---|---|---|---|
| 1. On a scale of 1 | to 5 where 1 is ve | ery difficult and 5 | is very easy, how eas | sy was the <b>set up</b> |
| and placement | of the PureWick <sup>TM</sup> | System? | | |
| 1 | 2 | 3 | 4 | 5 |
| 1 | 2 | 3 | т | 3 |
| Very difficult | Somewhat | Average | Somewhat easy | Very easy |
| • | difficult | difficulty | · | |
| | | , | | |
| Comments: | | | | |
| 2. On a scale of | 1 to 5 where 1 is | very difficult and | 5 is very easy, how ear | asy was |
| the <b>removal</b> of the PureWick <sup>TM</sup> FEC? | | | | |
| mo removar | or mic I wie Wiek | 120. | | |
| 1 | 2 | 3 | 4 | 5 |


| Very difficult | Somewhat<br>difficult | Average difficulty | Somewhat easy | Very easy |
|---|---|---|---|---|
| Comments: | | | | |
| 3. How would y sleep? | ou describe the dr | yness experience | ed with the PureWick <sup>7</sup> | <sup>TM</sup> System during |
| 1 | 2 3- 4 | | | |
| Never Dry (unacceptable) | | imes Dry<br>ceptable) | Usually Dry (acceptable) | Always Dry to<br>mostly always dry<br>(acceptable) |
| Comments: | , | - | | , |

# Appendix 15: Hollister® Female Urinary Pouch External Collection Device Participant Ease of use Questionnaire (Sample)

| Participant Number: | | Visit #: | Visit #: | |
|---|---|---|---|---|
| 1. On a scale of 1 to 5 where 1 is very difficult and 5 is very easy, how easy was the <b>placement</b> of the Hollister® Female Urinary Pouch External Collection Device? | | | | |
| 1 | 2 | 3 | 4 | 5 |
| Very difficult | Somewhat difficult | Average difficulty | Somewhat easy | Very easy |
| Comments: | | | | |
| 2. On a scale of 1 to 5 where 1 is very difficult and 5 is very easy, how easy was the <b>removal</b> of the Hollister® Female Urinary Pouch External Collection Device? | | | | |
| 1 | 2 | 3 | 4 | 5 |
| Very difficult | Somewhat difficult | Average difficulty | Somewhat easy | Very easy |
| Comments: | | | | |


| 1 | scribe the dryness experi<br>llection Device during sl | | ® Female Urinary |
|---|---|---|---|
| 1 | 2 | 3 | 4 |
| Never Dry<br>(unacceptable) | Sometimes Dry (unacceptable) | Usually Dry (acceptable) | Always Dry to<br>mostly always dry<br>(acceptable) |
| Comments: | | | • |

# **Appendix 16: End of Study Participant Preference Survey (Sample)**

| Thank you for participating in this study. Now that you have experienced the use of two urine collection devices, please answer a few questions about your experiences with the devices. As a reminder, during the study, you used two devices overnight while sleeping: During the first part of the study, you used the PureWick™ Urine Collection System/Hollister Female Urinary Pouch External Collection Device. During the second part of the study, you used the PureWick™ Urine Collection System/Hollister Female Urinary Pouch External Collection Device. | Participant Number: | |
|---|---|---|
| As a reminder, during the study, you used two devices overnight while sleeping: During the first part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection System/Hollister Female Urinary Pouch External Collection Device</i> . During the second part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection</i> | | |
| As a reminder, during the study, you used two devices overnight while sleeping: During the first part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection System/Hollister Female Urinary Pouch External Collection Device</i> . During the second part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection</i> | | |
| As a reminder, during the study, you used two devices overnight while sleeping: During the first part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection System/Hollister</i> Female Urinary Pouch External Collection Device. During the second part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection</i> | | |
| During the first part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection System/Hollister</i> Female Urinary Pouch External Collection Device. During the second part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection</i> | collection devices, please answer a few questions about your exp | eriences with the devices. |
| During the first part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection System/Hollister</i> Female Urinary Pouch External Collection Device. During the second part of the study, you used the <i>PureWick<sup>TM</sup> Urine Collection</i> | | |
| Female Urinary Pouch External Collection Device. During the second part of the study, you used the PureWick <sup>TM</sup> Urine Collection | As a reminder, during the study, you used two devices overnight | while sleeping: |
| | During the first part of the study, you used the $PureWick^{TM}$ $Urine Female$ $Urinary$ $Pouch$ $External$ $Collection$ $Device$ . | e Collection System/Hollister |
| | • • • • | |
| 1. Do you remember using each of these devices? | • | |
| Yes No | 1 33 | |

Ito
Ito
If No or if there is significant difficulty in differentiating the 2 study phases, discontinue the interview.>


| 2. | Which device did you prefer? PureWick™ Urine Collection System Hollister® Female Urinary Pouch External Collection Device |
|---|---|
| 3. | What made you choose the <purewick hollister=""> device? Why did you prefer that device?</purewick> |
| | <ask as="" better="" follow-up="" much="" participant's="" practical,="" preference="" questions,="" the="" to="" understand=""></ask> |
| 4. | Please think about how your skin felt when using each device. Which caused you to feel LESS skin irritation, the PureWick <sup>TM</sup> device or Hollister® device? PureWick <sup>TM</sup> Urine Collection System Hollister® Female Urinary Pouch External Collection Device No difference Do not recall |
| Why d | lid you choose the PureWick/Hollister? |

Thank you for taking the time to answer these questions!